CLINICAL TRIAL: NCT02453282
Title: A Phase III Randomized, Open-Label, Multi-Center, Global Study of MEDI4736 in Combination With Tremelimumab Therapy or MEDI4736 Monotherapy Versus Standard of Care Platinum-Based Chemotherapy in First Line Treatment of Patients With Advanced or Metastatic Non Small-Cell Lung Cancer (NSCLC)(MYSTIC).
Brief Title: Phase III Open Label First Line Therapy Study of MEDI 4736 (Durvalumab) With or Without Tremelimumab Versus SOC in Non Small-Cell Lung Cancer (NSCLC)
Acronym: MYSTIC
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D419AC00001; 2015-001279-39 (EudraCT Number)
Record Dates: First submitted 2015-05-20; First posted 2015-05-25 (Estimated); Results first posted 2019-11-29 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Non-Small-Cell Lung Carcinoma NSCLC
Keywords: NSCLC, PD-L1, MEDI4736, Tremelimumab, PFS, OS
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — durvalumab; CP protocol; Gemcitabine; Cisplatin; Carboplatin; Pemetrexed; tremelimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Monotherapy (Experimental): PD-L1 monoclonal Antibody monotherapy.
  Interventions: Biological: MEDI4736 (Durvalumab)
- Combination Therapy (Experimental): PD-L1+Tremelimumab combination therapy
  Interventions: Biological: MEDI4736 (Durvalumab)+Tremelimumab; Biological: Tremelimumab
- Standard of Care (Active Comparator): Standard of Care chemotherapy treatment
  Interventions: Drug: Paclitaxel + Carboplatin; Drug: Gemcitabine + Cisplatin; Drug: Gemcitabine + Carboplatin; Drug: Pemetrexed + Cisplatin; Drug: Pemetrexed + Carboplatin

INTERVENTIONS:
Biological: MEDI4736 (Durvalumab)
  Arms: Monotherapy
Biological: MEDI4736 (Durvalumab)+Tremelimumab
  Arms: Combination Therapy
Drug: Paclitaxel + Carboplatin — Chemotherapy Agents
  Other Names: Platinum based Standard of Care Chemotherapy
  Arms: Standard of Care
Drug: Gemcitabine + Cisplatin — Chemotherapy Agents
  Other Names: Platinum based Standard of Care Chemotherapy
  Arms: Standard of Care
Drug: Gemcitabine + Carboplatin — Chemotherapy Agents
  Other Names: Platinum based Standard of Care Chemotherapy
  Arms: Standard of Care
Drug: Pemetrexed + Cisplatin — Chemotherapy Agents
  Other Names: Platinum based Standard of Care Chemotherapy
  Arms: Standard of Care
Drug: Pemetrexed + Carboplatin — Chemotherapy Agents
  Other Names: Platinum based Standard of Care Chemotherapy
  Arms: Standard of Care
Biological: Tremelimumab
  Arms: Combination Therapy

SUMMARY:
This is a randomized, open-label, multi-center, global, Phase III study to determine the efficacy and safety of MEDI4736 + tremelimumab combination therapy and MEDI4736 monotherapy versus platinum-based SoC chemotherapy in the first-line treatment of patients with epidermal growth factor receptor (EGFR) and anaplastic lymphoma kinase (ALK) wild-type locally advanced or metastatic NSCLC

DETAILED DESCRIPTION:
Patients will be randomized in a 1:1:1 ratio to receive treatment with MEDI4736 + tremelimumab combination therapy, MEDI4736 monotherapy, or Standard of Care (SoC) therapy.

ELIGIBILITY:
Inclusion Criteria:

For inclusion in the study, patients should fulfill the following criteria:

* Aged at least 18 years
* Documented evidence of Stage IV NSCLC
* No sensitizing EGFR mutation or ALK rearrangement
* No prior chemotherapy or any other systemic therapy for recurrent/metastatic NSCLC
* World Health Organization (WHO) Performance Status of 0 or 1

Exclusion Criteria:

Patients should not enter the study if any of the following exclusion criteria are fulfilled:

1. Mixed small-cell lung cancer and NSCLC histology, sarcomatoid variant
2. Brain metastases or spinal cord compression unless asymptomatic, treated and stable (not requiring steroids)
3. Prior exposure to Immunomodulatory therapy (IMT), including, but not limited to, other anti-cytotoxic T-lymphocyte-associated antigen 4 (CTLA-4), anti-programmed cell death1 (PD-1), anti-programmed cell death ligand 1 (PD-L1), or anti PD-L2 antibodies, excluding therapeutic anticancer vaccines
4. Active or prior documented autoimmune or inflammatory disorders (including inflammatory bowel disease [eg, colitis or Crohn's disease]

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1118 (Actual)
Dates: Start 2015-07-21 (Actual); Primary Completion 2018-10-04 (Actual); Study Completion 2025-12-31 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Stuart McIntosh, MD, Study Director — AstraZeneca, Alderley Park, Cheshire, UK; Naiyer Rizvi, MD, Principal Investigator — Columbia University Medical Center, New York, NY, USA
Locations (164):
- United States (31):
  - Research Site, Scottsdale, Arizona
  - Research Site, Tucson, Arizona
  - Research Site, Yuma, Arizona
  - Research Site, Bakersfield, California
  - Research Site, Fullerton, California
  - Research Site, La Jolla, California
  - Research Site, Los Angeles, California
  - Research Site, Redondo Beach, California
  - Research Site, Sacramento, California
  - Research Site, San Luis Obispo, California
  - Research Site, Santa Maria, California
  - Research Site, West Hollywood, California
  - Research Site, New Haven, Connecticut
  - Research Site, Jacksonville, Florida
  - Research Site, Pembroke Pines, Florida
  - Research Site, Tampa, Florida
  - Research Site, Athens, Georgia
  - Research Site, Honolulu, Hawaii
  - Research Site, Baltimore, Maryland
  - Research Site, Minneapolis, Minnesota
  - Research Site, St Louis, Missouri
  - Research Site, Omaha, Nebraska
  - Research Site, Summit, New Jersey
  - Research Site, Mineola, New York
  - Research Site, New York, New York
  - Research Site, Charlotte, North Carolina
  - Research Site, Cleveland, Ohio
  - Research Site, North Charleston, South Carolina
  - Research Site, Nashville, Tennessee
  - Research Site, Richmond, Virginia
  - Research Site, Madison, Wisconsin
- Australia (7):
  - Research Site, Box Hill
  - Research Site, Gosford
  - Research Site, Kogarah
  - Research Site, Melbourne
  - Research Site, Port Macquarie
  - Research Site, Southport
  - Research Site, St Leonards
- Belgium (5):
  - Research Site, Brussels
  - Research Site, Charleroi
  - Research Site, Duffel
  - Research Site, Leuven
  - Research Site, Liège
- Canada (9):
  - Research Site, Greater Sudbury, Ontario
  - Research Site, Kingston, Ontario
  - Research Site, Newmarket, Ontario
  - Research Site, Oshawa, Ontario
  - Research Site, Sault Ste. Marie, Ontario
  - Research Site, St. Catharines, Ontario
  - Research Site, Toronto, Ontario
  - Research Site, Regina, Saskatchewan
  - Research Site, Saskatoon, Saskatchewan
- France (6):
  - Research Site, Bordeaux
  - Research Site, Brest
  - Research Site, Créteil
  - Research Site, Lille
  - Research Site, Lyon
  - Research Site, Marseille
- Germany (18):
  - Research Site, Aachen
  - Research Site, Bad Berka
  - Research Site, Berlin
  - Research Site, Freiburg im Breisgau
  - Research Site, Gauting
  - Research Site, Hamburg
  - Research Site, Heidelberg
  - Research Site, Hemer
  - Research Site, Homburg/Saar
  - Research Site, Immenhausen
  - Research Site, Löwenstein
  - Research Site, Lübeck
  - Research Site, Mainz
  - Research Site, Münster
  - Research Site, Oldenburg
  - Research Site, Ulm
  - Research Site, Velbert
  - Research Site, Würzburg
- Hungary (9):
  - Research Site, Budapest
  - Research Site, Deszk
  - Research Site, Edelény
  - Research Site, Kaposvár
  - Research Site, Kecskemét
  - Research Site, Miskolc
  - Research Site, Nyíregyháza
  - Research Site, Pécs
  - Research Site, Székesfehérvár
- Italy (5):
  - Research Site, Genova
  - Research Site, Meldola
  - Research Site, Milan
  - Research Site, San Giovanni Rotondo
  - Research Site, Siena
- Japan (27):
  - Research Site, Fukushima
  - Research Site, Himeji-shi
  - Research Site, Hirakata-shi
  - Research Site, Hirosaki-shi
  - Research Site, Iizuka-shi
  - Research Site, Iwakuni-shi
  - Research Site, Izumi-shi
  - Research Site, Kanazawa
  - Research Site, Kishiwada-shi
  - Research Site, Kobe
  - Research Site, Koga-shi
  - Research Site, Kyoto
  - Research Site, Mitaka-shi
  - Research Site, Nagaoka-shi
  - Research Site, Nagoya
  - Research Site, Okayama
  - Research Site, Osaka
  - Research Site, Saga
  - Research Site, Saitama-shi
  - Research Site, Sakaishi
  - Research Site, Sayama
  - Research Site, Sendai
  - Research Site, Shinjuku-ku
  - Research Site, Tokushima
  - Research Site, Ube-shi
  - Research Site, Yokohama
  - Research Site, Yokosuka-shi
- Netherlands (7):
  - Research Site, 's-Hertogenbosch
  - Research Site, Amsterdam
  - Research Site, Arnhem
  - Research Site, Breda
  - Research Site, Groningen
  - Research Site, Maastricht
  - Research Site, Rotterdam
- Russia (4):
  - Research Site, Moscow
  - Research Site, Obninsk
  - Research Site, Omsk
  - Research Site, Saint Petersburg
- South Korea (12):
  - Research Site, Busan
  - Research Site, Changwon-si
  - Research Site, Cheongju-si
  - Research Site, Daegu
  - Research Site, Daejeon
  - Research Site, Goyang-si
  - Research Site, Incheon
  - Research Site, Jinju
  - Research Site, Seongnam-si
  - Research Site, Seoul
  - Research Site, Suwon
  - Research Site, Ulsan
- Spain (11):
  - Research Site, A Coruña
  - Research Site, Alicante
  - Research Site, Barcelona
  - Research Site, Girona
  - Research Site, Jaén
  - Research Site, León
  - Research Site, Madrid
  - Research Site, Majadahonda
  - Research Site, Málaga
  - Research Site, Seville
  - Research Site, Valencia
- Switzerland (2):
  - Research Site, Bellinzona
  - Research Site, Lausanne
- Taiwan (5):
  - Research Site, Kaohsiung City
  - Research Site, Taichung
  - Research Site, Tainan
  - Research Site, Taipei
  - Research Site, Taoyuan District
- Thailand (4):
  - Research Site, Bangkok
  - Research Site, Chiang Mai
  - Research Site, Hat Yai
  - Research Site, Khon Kaen
- Vietnam (2):
  - Research Site, Hanoi
  - Research Site, Ho Chi Minh City

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- [Derived] Garon EB, Cho BC, Reinmuth N, Lee KH, Luft A, Ahn MJ, Robinet G, Le Moulec S, Natale R, Schneider J, Shepherd FA, Garassino MC, Geater SL, Szekely ZP, Van Ngoc T, Liu F, Scheuring U, Patel N, Peters S, Rizvi NA. Patient-Reported Outcomes with Durvalumab With or Without Tremelimumab Versus Standard Chemotherapy as First-Line Treatment of Metastatic Non-Small-Cell Lung Cancer (MYSTIC). Clin Lung Cancer. 2021 Jul;22(4):301-312.e8. doi: 10.1016/j.cllc.2021.02.010. Epub 2021 Feb 19. PMID 33775558
- [Derived] Rizvi NA, Cho BC, Reinmuth N, Lee KH, Luft A, Ahn MJ, van den Heuvel MM, Cobo M, Vicente D, Smolin A, Moiseyenko V, Antonia SJ, Le Moulec S, Robinet G, Natale R, Schneider J, Shepherd FA, Geater SL, Garon EB, Kim ES, Goldberg SB, Nakagawa K, Raja R, Higgs BW, Boothman AM, Zhao L, Scheuring U, Stockman PK, Chand VK, Peters S; MYSTIC Investigators. Durvalumab With or Without Tremelimumab vs Standard Chemotherapy in First-line Treatment of Metastatic Non-Small Cell Lung Cancer: The MYSTIC Phase 3 Randomized Clinical Trial. JAMA Oncol. 2020 May 1;6(5):661-674. doi: 10.1001/jamaoncol.2020.0237. PMID 32271377
- See also: Related Info — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D419AC00001&attachmentIdentifier=44a72f97-af1b-4e4c-8b0e-d65a6cc9cc88&fileName=D419AC00001_Statistical_Analysis_Plan_Redacted.pdf&versionIdentifier=
- See also: Related Info — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D419AC00001&attachmentIdentifier=cbfa257d-1cad-4287-aa97-aaad910d92df&fileName=D419AC00001_Version_8.0_CSP_Redacted.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 194 centers across 17 countries in Asia, Australia, Europe and North America randomized adults with epidermal growth factor receptor and anaplastic lymphoma kinase wild-type advanced or metastatic non-small cell lung cancer in this study. First participant was randomized on 14 August 2015 and final data cut-off date was 04 October 2018.
Pre-assignment Details: A total of 1118 participants were randomized in a 1:1:1 ratio in stratified manner as per programmed cell death ligand 1 (PD-L1) tumor expression status (PD-L1 [tumor cell (TC) >=25%] versus (Vs) PD-L1 [TC <25%]) and histology (squamous Vs non-squamous) to receive durvalumab alone, durvalumab + tremelimumab, or standard of care (SoC) chemotherapy.
Groups:
- Durvalumab Monotherapy: Participants received durvalumab 20 milligram per kilogram (mg/kg) intravenous (IV) infusion every 4 weeks (Q4W) until worsening of the disease under investigation, unless specific treatment discontinuation criteria were met.
- Durvalumab + Tremelimumab: Participants received durvalumab 20 mg/kg and tremelimumab 1 mg/kg IV infusion Q4W in combination for up to 4 doses/cycles. Participants then continued on durvalumab 20 mg/kg Q4W, starting on Week 16 until worsening of the disease under investigation, unless specific treatment discontinuation criteria were met.
- SoC Chemotherapy: Participants received 1 of the following IV infusion treatment combinations on Day 1 of each 21-day cycle for 4 to 6 cycles or until worsening of disease under investigation, unless specific treatment discontinuation criteria were met.
  1. Paclitaxel 200 mg/square meter (m^2) and carboplatin area under the plasma drug concentration-time curve (AUC) 5 or 6 mg*minute per milliliter (mg*min/mL).
  2. Gemcitabine 1000 or 1250 mg/m^2 and cisplatin 75 or 80 mg/m^2. Additional dose of Gemcitabine 1000 or 1250 mg/m^2 on Day 8 of each cycle (For squamous tumors only).
  3. Gemcitabine 1000 or 1250 mg/m^2 and carboplatin AUC 5 or 6 mg*min/mL. Additional dose of Gemcitabine 1000 or 1250 mg/m^2 on Day 8 of each cycle (For squamous tumors only).
  4. Pemetrexed 500 mg/m^2 and cisplatin 75 mg/m^2 (For non-squamous tumors only; pemetrexed maintenance dose was permitted).
  5. Pemetrexed 500 mg/m^2 and carboplatin AUC 5 or 6 mg*min/mL (For non-squamous tumors only; pemetrexed maintenance dose was permitted).
Period: Overall Study
Arm/Group | Durvalumab Monotherapy | Durvalumab + Tremelimumab | SoC Chemotherapy
Started | 374 | 372 | 372
Received Treatment | 369 | 371 | 352
Completed | 0 | 0 | 0
Not Completed | 374 | 372 | 372
Not completed — Death | 275 | 277 | 296
Not completed — Lost to Follow-up | 1 | 0 | 2
Not completed — Withdrawal by Subject | 12 | 10 | 11
Not completed — Participants ongoing at data cut-off | 85 | 84 | 62
Not completed — Other | 1 | 1 | 1

BASELINE CHARACTERISTICS:
Population: Full analysis set (FAS) included all randomized participants analyzed on an intent-to-treat (ITT) basis.
Groups:
- Durvalumab Monotherapy: Participants received durvalumab 20 mg/kg IV infusion Q4W until worsening of the disease under investigation, unless specific treatment discontinuation criteria were met.
- SoC Chemotherapy: Participants received 1 of the following IV infusion treatment combinations on Day 1 of each 21-day cycle for 4 to 6 cycles or until worsening of disease under investigation, unless specific treatment discontinuation criteria were met.
  1. Paclitaxel 200 mg/m^2 and carboplatin AUC 5 or 6 mg*min/mL.
  2. Gemcitabine 1000 or 1250 mg/m^2 and cisplatin 75 or 80 mg/m^2. Additional dose of Gemcitabine 1000 or 1250 mg/m^2 on Day 8 of each cycle (For squamous tumors only).
  3. Gemcitabine 1000 or 1250 mg/m^2 and carboplatin AUC 5 or 6 mg*min/mL. Additional dose of Gemcitabine 1000 or 1250 mg/m^2 on Day 8 of each cycle (For squamous tumors only).
  4. Pemetrexed 500 mg/m^2 and cisplatin 75 mg/m^2 (For non-squamous tumors only; pemetrexed maintenance dose was permitted).
  5. Pemetrexed 500 mg/m^2 and carboplatin AUC 5 or 6 mg*min/mL (For non-squamous tumors only; pemetrexed maintenance dose was permitted).
- Total: Total of all reporting groups
Arm/Group | Durvalumab Monotherapy | Durvalumab + Tremelimumab | SoC Chemotherapy | Total
Number analyzed (Participants) | 374 | 372 | 372 | 1118
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.2 (10.30) | 64.3 (9.52) | 63.6 (9.36) | 63.7 (9.74)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 118 | 106 | 122 | 346
  Male | 256 | 266 | 250 | 772
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 15 | 13 | 6 | 34
  Not Hispanic or Latino | 359 | 358 | 366 | 1083
  Unknown or Not Reported | 0 | 1 | 0 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 243 | 249 | 243 | 735
  Black or African American | 3 | 3 | 4 | 10
  Asian | 125 | 118 | 120 | 363
  Native Hawaiian or other Pacific Islander | 0 | 0 | 2 | 2
  Other | 3 | 1 | 3 | 7
  Missing | 0 | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (OS); PD-L1 (TC >=25%) Analysis Set Population, Durvalumab Monotherapy Vs SoC Chemotherapy and Durvalumab + Tremelimumab Vs SoC Chemotherapy
Description: The OS was defined as the time from the date of randomization until death due to any cause (ie, date of death or censoring - date of randomization + 1). Any participant not known to have died at the time of analysis were censored based on the last recorded date on which the participant was known to be alive. Median OS was calculated using the Kaplan-Meier technique.
Time Frame: From baseline (Day 1, Week 0) until death due to any cause, assessed up to the data cut-off date (a maximum of approximately 3 years).
Population: The PD-L1 (TC >=25%) analysis set included subset of participants in the FAS whose PD-L1 status was PD-L1 (TC >=25%) as defined by Ventana PD-L1 (SP263) assay (ie, >=25% TCs expressing PD-L1 on the membrane). Comparison of durvalumab monotherapy Vs SoC and durvalumab + tremelimumab Vs SoC reporting groups were analysed for primary outcome measure.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Durvalumab Monotherapy | Durvalumab + Tremelimumab | SoC Chemotherapy
Number analyzed (Participants) | 163 | 163 | 162
months | 16.3 [12.2 to 20.8] | 11.9 [9.0 to 17.7] | 12.9 [10.5 to 15.0]
Statistical Analysis 1: Comparison: Durvalumab Monotherapy vs SoC Chemotherapy; Durvalumab Monotherapy Vs SoC Chemotherapy; Test type: Superiority; p = 0.036, Log Rank — The 2-sided p-value was calculated using a stratified log-rank test adjusting for histology (squamous Vs non-squamous), with ties handled by the Breslow approach; Hazard Ratio (HR) = 0.76, 97.54% CI 2-sided [0.564 to 1.019] — The HR and confidence interval (CI) were calculated using a stratified Cox proportional hazards model, adjusting for histology (squamous Vs non-squamous), with ties handled by the Breslow approach
Statistical Analysis 2: Comparison: Durvalumab + Tremelimumab vs SoC Chemotherapy; Durvalumab + Tremelimumab Vs SoC Chemotherapy; Test type: Superiority; p = 0.202, Log Rank — [p-value comment as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.85, 98.77% CI 2-sided [0.611 to 1.173] — The HR and CI were calculated using a stratified Cox proportional hazards model, adjusting for histology (squamous Vs non-squamous), with ties handled by the Breslow approach

2. Primary Outcome: Progression-Free Survival (PFS); PD-L1 (TC >=25%) Analysis Set Population, Durvalumab + Tremelimumab Vs SoC Chemotherapy
Description: The PFS per Response Evaluation Criteria in Solid Tumors, version 1.1 (RECIST 1.1) using blinded independent central review (BICR) assessments was defined as the time from the date of randomization until the date of objective disease progression or death (by any cause in the absence of progression) regardless of whether the participant withdraw from randomized therapy or received another anti-cancer therapy prior to progression (ie, date of PFS event or censoring - date of randomization + 1). Progressive disease (PD) was defined as at least a 20% increase in the sum of diameters of target lesions (TLs) and an absolute increase of at least 5 millimeter (mm), taking as reference the smallest sum of diameters since treatment started including the baseline sum of diameters. Median PFS was calculated using the Kaplan-Meier technique.
Time Frame: Tumour scans performed at baseline then every 6 weeks up to 48 weeks relative to the date of randomization, then every 8 weeks thereafter until confirmed disease progression. Assessed up to the data cut-off date (a maximum of approximately 3 years).
Population: The PD-L1 (TC >=25%) analysis set included the subset of participants in the FAS whose PD-L1 status was PD-L1 (TC >=25%) as defined by the Ventana PD-L1 (SP263) assay (ie, >=25% TCs expressing PD-L1 on the membrane). Comparison of durvalumab + tremelimumab Vs SoC chemotherapy reporting groups were analysed for the primary outcome measure.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Durvalumab + Tremelimumab | SoC Chemotherapy
Number analyzed (Participants) | 163 | 162
months | 3.9 [2.8 to 5.0] | 5.4 [4.6 to 5.8]
Statistical Analysis 1: Comparison: Durvalumab + Tremelimumab vs SoC Chemotherapy; Durvalumab + Tremelimumab Vs SoC Chemotherapy; Test type: Superiority; p = 0.705, Log Rank — The analysis was performed using stratified log-rank test adjusting for histology (squamous Vs non-squamous), with ties handled by the Breslow approach; Hazard Ratio (HR) = 1.05, 99.5% CI 2-sided [0.722 to 1.534] — [estimate comment as in outcome 1, analysis 2]

3. Secondary Outcome: OS; PD-L1 (TC >=25%) Analysis Set Population, Durvalumab + Tremelimumab Vs Durvalumab Monotherapy
Description: as for outcome 1
Time Frame: From baseline until death due to any cause, assessed up to the data cut-off date (a maximum of approximately 3 years).
Population: The PD-L1 (TC >=25%) analysis set included the subset of participants in the FAS whose PD-L1 status was PD-L1 (TC >=25%) as defined by the Ventana PD-L1 (SP263) assay (ie, >=25% TCs expressing PD-L1 on the membrane). Comparison of durvalumab + tremelimumab Vs durvalumab monotherapy reporting groups were analysed for the secondary outcome measure.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Durvalumab Monotherapy | Durvalumab + Tremelimumab | SoC Chemotherapy
Number analyzed (Participants) | 163 | 163 | 162
months | 16.3 [12.2 to 20.8] | 11.9 [9.0 to 17.7] | 12.9 [10.5 to 15.0]
Statistical Analysis 1: Comparison: Durvalumab Monotherapy vs Durvalumab + Tremelimumab; Durvalumab + Tremelimumab Vs Durvalumab Monotherapy; Test type: Superiority; p = 0.523, Log Rank — [p-value comment as in outcome 1, analysis 1]; Hazard Ratio (HR) = 1.09, 95% CI 2-sided [0.836 to 1.421] — [estimate comment as in outcome 1, analysis 2]

4. Secondary Outcome: OS; PD-L1 (TC >=1%) Analysis Set Population
Description: as for outcome 1
Time Frame: From baseline until death due to any cause, assessed up to the data cut-off date (a maximum of approximately 3 years).
Population: The PD-L1 (TC >=1%) analysis set included the subset of participants in the FAS whose PD-L1 status is PD-L1 (TC >=1%) as defined by the Ventana PD-L1 (SP263) assay (ie, >=1% TC expressing PD-L1 on the membrane).
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Durvalumab Monotherapy | Durvalumab + Tremelimumab | SoC Chemotherapy
Number analyzed (Participants) | 279 | 296 | 289
months | 14.6 [10.5 to 17.7] | 10.9 [9.1 to 13.5] | 12.3 [10.6 to 14.6]
Statistical Analysis 1: Comparison: Durvalumab Monotherapy vs SoC Chemotherapy; Durvalumab Monotherapy Vs SoC Chemotherapy; Test type: Superiority; p = 0.194, Log Rank — The 2-sided p-value was calculated using a stratified log-rank test adjusting for PD-L1 status (>=25% Vs <25%) and histology (squamous Vs non-squamous), with ties handled by the Breslow approach; Hazard Ratio (HR) = 0.88, 95% CI 2-sided [0.725 to 1.067] — The HR and CI were calculated using a stratified Cox proportional hazards model, adjusting for PD-L1 status (>=25% Vs <25%) and histology (squamous Vs non-squamous), with ties handled by the Breslow approach
Statistical Analysis 2: Comparison: Durvalumab + Tremelimumab vs SoC Chemotherapy; Durvalumab + Tremelimumab Vs SoC Chemotherapy; Test type: Superiority; p = 0.952, Log Rank — [p-value comment as in outcome 4, analysis 1]; Hazard Ratio (HR) = 1.01, 95% CI 2-sided [0.834 to 1.213] — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 3: Comparison: Durvalumab Monotherapy vs Durvalumab + Tremelimumab; Durvalumab + Tremelimumab Vs Durvalumab Monotherapy; Test type: Superiority; p = 0.218, Log Rank — [p-value comment as in outcome 4, analysis 1]; Hazard Ratio (HR) = 1.13, 95% CI 2-sided [0.931 to 1.371] — [estimate comment as in outcome 4, analysis 1]

5. Secondary Outcome: OS; FAS Population
Description: as for outcome 1
Time Frame: From baseline until death due to any cause, assessed up to the data cut-off date (a maximum of approximately 3 years).
Population: The FAS included all randomized participants analyzed on an ITT basis.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Durvalumab Monotherapy | Durvalumab + Tremelimumab | SoC Chemotherapy
Number analyzed (Participants) | 374 | 372 | 372
months | 12.3 [10.1 to 14.9] | 11.2 [9.5 to 12.9] | 11.8 [10.5 to 13.3]
Statistical Analysis 1: Comparison: Durvalumab Monotherapy vs SoC Chemotherapy; Durvalumab Monotherapy Vs SoC Chemotherapy; Test type: Superiority; p = 0.602, Log Rank — [p-value comment as in outcome 4, analysis 1]; Hazard Ratio (HR) = 0.96, 95% CI 2-sided [0.812 to 1.128] — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 2: Comparison: Durvalumab + Tremelimumab vs SoC Chemotherapy; Durvalumab + Tremelimumab Vs SoC Chemotherapy; Test type: Superiority; p = 0.430, Log Rank — [p-value comment as in outcome 4, analysis 1]; Hazard Ratio (HR) = 0.94, 95% CI 2-sided [0.794 to 1.103] — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 3: Comparison: Durvalumab Monotherapy vs Durvalumab + Tremelimumab; Durvalumab + Tremelimumab Vs Durvalumab Monotherapy; Test type: Superiority; p = 0.802, Log Rank — [p-value comment as in outcome 4, analysis 1]; Hazard Ratio (HR) = 0.98, 95% CI 2-sided [0.828 to 1.157] — [estimate comment as in outcome 4, analysis 1]

6. Secondary Outcome: PFS; PD-L1 (TC >=25%) Analysis Set Population, Durvalumab Monotherapy Vs SoC Chemotherapy and Durvalumab + Tremelimumab Vs Durvalumab Monotherapy
Description: The PFS per RECIST 1.1 using BICR assessments was defined as the time from the date of randomization until the date of objective disease progression or death (by any cause in the absence of progression) regardless of whether the participant withdraw from randomized therapy or received another anti-cancer therapy prior to progression (ie, date of PFS event or censoring - date of randomization + 1). The PD was defined as at least a 20% increase in the sum of diameters of TLs and an absolute increase of at least 5 mm, taking as reference the smallest sum of diameters since treatment started including the baseline sum of diameters. Median PFS was calculated using the Kaplan-Meier technique.
Time Frame: as for outcome 2
Population: The PD-L1 (TC >=25%) analysis set included subset of participants in the FAS whose PD-L1 status was PD-L1 (TC >=25%) as defined by Ventana PD-L1 (SP263) assay (ie, >=25% TCs expressing PD-L1 on the membrane). Comparison of durvalumab + tremelimumab Vs durvalumab and durvalumab Vs SoC reporting groups were analysed for secondary outcome measure.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Durvalumab Monotherapy | Durvalumab + Tremelimumab | SoC Chemotherapy
Number analyzed (Participants) | 163 | 163 | 162
months | 4.7 [3.1 to 6.3] | 3.9 [2.8 to 5.0] | 5.4 [4.6 to 5.8]
Statistical Analysis 1: Comparison: Durvalumab Monotherapy vs SoC Chemotherapy; Durvalumab Monotherapy Vs SoC Chemotherapy; Test type: Superiority; p = 0.324, Log Rank — [p-value comment as in outcome 2, analysis 1]; Hazard Ratio (HR) = 0.87, 95% CI 2-sided [0.667 to 1.143] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 2: Comparison: Durvalumab Monotherapy vs Durvalumab + Tremelimumab; Durvalumab + Tremelimumab Vs Durvalumab Monotherapy; Test type: Superiority; p = 0.207, Log Rank — [p-value comment as in outcome 2, analysis 1]; Hazard Ratio (HR) = 1.18, 95% CI 2-sided [0.911 to 1.541] — [estimate comment as in outcome 1, analysis 2]

7. Secondary Outcome: PFS; PD-L1 (TC >=1%) Analysis Set Population
Description: as for outcome 6
Time Frame: as for outcome 2
Population: as for outcome 4
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Durvalumab Monotherapy | Durvalumab + Tremelimumab | SoC Chemotherapy
Number analyzed (Participants) | 279 | 296 | 289
months | 3.6 [2.8 to 4.2] | 2.8 [2.5 to 3.4] | 5.5 [4.9 to 5.7]
Statistical Analysis 1: Comparison: Durvalumab Monotherapy vs SoC Chemotherapy; Durvalumab Monotherapy Vs SoC Chemotherapy; Test type: Superiority; p = 0.383, Log Rank — The analysis was performed using stratified log-rank test adjusting for PD-L1 status (>=25% Vs <25%) and histology (squamous Vs non-squamous), with ties handled by the Breslow approach; Hazard Ratio (HR) = 1.09, 95% CI 2-sided [0.894 to 1.339] — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 2: Comparison: Durvalumab + Tremelimumab vs SoC Chemotherapy; Durvalumab + Tremelimumab Vs SoC Chemotherapy; Test type: Superiority; p = 0.001, Log Rank — [p-value comment as in outcome 7, analysis 1]; Hazard Ratio (HR) = 1.38, 95% CI 2-sided [1.136 to 1.678] — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 3: Comparison: Durvalumab Monotherapy vs Durvalumab + Tremelimumab; Durvalumab + Tremelimumab Vs Durvalumab Monotherapy; Test type: Superiority; p = 0.138, Log Rank — [p-value comment as in outcome 7, analysis 1]; Hazard Ratio (HR) = 1.16, 95% CI 2-sided [0.954 to 1.403] — [estimate comment as in outcome 4, analysis 1]

8. Secondary Outcome: PFS; FAS Population
Description: as for outcome 6
Time Frame: as for outcome 2
Population: The FAS included all randomized participants analyzed on an ITT basis.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Durvalumab Monotherapy | Durvalumab + Tremelimumab | SoC Chemotherapy
Number analyzed (Participants) | 374 | 372 | 372
months | 2.8 [2.6 to 3.1] | 2.9 [2.6 to 3.4] | 5.4 [4.8 to 5.6]
Statistical Analysis 1: Comparison: Durvalumab Monotherapy vs SoC Chemotherapy; Durvalumab Monotherapy Vs SoC Chemotherapy; Test type: Superiority; p = 0.015, Log Rank — [p-value comment as in outcome 7, analysis 1]; Hazard Ratio (HR) = 1.24, 95% CI 2-sided [1.043 to 1.475] — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 2: Comparison: Durvalumab + Tremelimumab vs SoC Chemotherapy; Durvalumab + Tremelimumab Vs SoC Chemotherapy; Test type: Superiority; p = 0.010, Log Rank — [p-value comment as in outcome 7, analysis 1]; Hazard Ratio (HR) = 1.25, 95% CI 2-sided [1.054 to 1.485] — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 3: Comparison: Durvalumab Monotherapy vs Durvalumab + Tremelimumab; Durvalumab + Tremelimumab Vs Durvalumab Monotherapy; Test type: Superiority; p = 0.984, Log Rank — [p-value comment as in outcome 7, analysis 1]; Hazard Ratio (HR) = 1.00, 95% CI 2-sided [0.845 to 1.179] — [estimate comment as in outcome 4, analysis 1]

9. Secondary Outcome: Objective Response Rate (ORR); PD-L1 (TC >=25%) Analysis Set Population
Description: The ORR per RECIST 1.1 using BICR assessments was defined as the percentage of participants with at least 1 visit response of Complete Response (CR) or Partial Response (PR). The CR was defined as disappearance of all TLs (any pathological lymph nodes selected as TLs must have a reduction in short axis to <10 mm) and PR was defined as at least a 30% decrease in the sum of diameters of TLs (taking as reference the baseline sum of diameters as long as criteria for PD are not met).
Time Frame: as for outcome 2
Population: The PD-L1 (TC >=25%) analysis set included the subset of participants in the FAS whose PD-L1 status was PD-L1 (TC >=25%) as defined by the Ventana PD-L1 (SP263) assay (ie, >=25% TC expressing PD-L1 on the membrane).
Measure: Number; unit: percentage of participants
Arm/Group | Durvalumab Monotherapy | Durvalumab + Tremelimumab | SoC Chemotherapy
Number analyzed (Participants) | 163 | 163 | 162
percentage of participants | 35.6 | 34.4 | 37.7
Statistical Analysis 1: Comparison: Durvalumab Monotherapy vs SoC Chemotherapy; Durvalumab Monotherapy Vs SoC Chemotherapy; Test type: Superiority; p = 0.698, Regression, Logistic — P-value is based on twice the change in log-likelihood resulting from the addition of a treatment factor to the model; Odds Ratio (OR) = 0.91, 95% CI 2-sided [0.582 to 1.437] — The analysis was performed using logistic regression adjusting for histology (squamous Vs non-squamous), with 95% CI calculated by profile likelihood
Statistical Analysis 2: Comparison: Durvalumab + Tremelimumab vs SoC Chemotherapy; Durvalumab + Tremelimumab Vs SoC Chemotherapy; Test type: Superiority; p = 0.534, Regression, Logistic — P-value is based on twice the change in log-likelihood resulting from the addition of a treatment factor to the model; Odds Ratio (OR) = 0.87, 95% CI 2-sided [0.549 to 1.363] — [estimate comment as in outcome 9, analysis 1]
Statistical Analysis 3: Comparison: Durvalumab Monotherapy vs Durvalumab + Tremelimumab; Durvalumab + Tremelimumab Vs Durvalumab Monotherapy; Test type: Superiority; p = 0.820, Regression, Logistic — P-value is based on twice the change in log-likelihood resulting from the addition of a treatment factor to the model; Odds Ratio (OR) = 0.95, 95% CI 2-sided [0.601 to 1.496] — [estimate comment as in outcome 9, analysis 1]

10. Secondary Outcome: ORR; PD-L1 (TC >=1%) Analysis Set Population
Description: The ORR per RECIST 1.1 using BICR assessments was defined as the percentage of participants with at least 1 visit response of CR or PR. The CR was defined as disappearance of all TLs (any pathological lymph nodes selected as TLs must have a reduction in short axis to <10 mm) and PR was defined as at least a 30% decrease in the sum of diameters of TLs (taking as reference the baseline sum of diameters as long as criteria for PD are not met).
Time Frame: as for outcome 2
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | Durvalumab Monotherapy | Durvalumab + Tremelimumab | SoC Chemotherapy
Number analyzed (Participants) | 279 | 296 | 289
percentage of participants | 26.5 | 25.3 | 33.6
Statistical Analysis 1: Comparison: Durvalumab Monotherapy vs SoC Chemotherapy; Durvalumab Monotherapy Vs SoC Chemotherapy; Test type: Superiority; p = 0.050, Regression, Logistic — P-value is based on twice the change in log-likelihood resulting from the addition of a treatment factor to the model; Odds Ratio (OR) = 0.69, 95% CI 2-sided [0.480 to 1.000] — The analysis was performed using logistic regression adjusting for histology (squamous Vs non squamous) and PD-L1 status (>=25% Vs <25%), with 95% CI calculated by profile likelihood
Statistical Analysis 2: Comparison: Durvalumab + Tremelimumab vs SoC Chemotherapy; Durvalumab + Tremelimumab Vs SoC Chemotherapy; Test type: Superiority; p = 0.029, Regression, Logistic — P-value is based on twice the change in log-likelihood resulting from the addition of a treatment factor to the model; Odds Ratio (OR) = 0.67, 95% CI 2-sided [0.464 to 0.959] — [estimate comment as in outcome 10, analysis 1]
Statistical Analysis 3: Comparison: Durvalumab Monotherapy vs Durvalumab + Tremelimumab; Durvalumab + Tremelimumab Vs Durvalumab Monotherapy; Test type: Superiority; p = 0.887, Regression, Logistic — P-value is based on twice the change in log-likelihood resulting from the addition of a treatment factor to the model; Odds Ratio (OR) = 0.97, 95% CI 2-sided [0.661 to 1.430] — [estimate comment as in outcome 10, analysis 1]

11. Secondary Outcome: ORR; FAS Population
Description: as for outcome 10
Time Frame: as for outcome 2
Population: The FAS included all randomized participants analyzed on an ITT basis.
Measure: Number; unit: percentage of participants
Arm/Group | Durvalumab Monotherapy | Durvalumab + Tremelimumab | SoC Chemotherapy
Number analyzed (Participants) | 374 | 372 | 372
percentage of participants | 22.2 | 24.7 | 30.1
Statistical Analysis 1: Comparison: Durvalumab Monotherapy vs SoC Chemotherapy; Durvalumab Monotherapy Vs SoC Chemotherapy; Test type: Superiority; p = 0.012, Regression, Logistic — P-value is based on twice the change in log-likelihood resulting from the addition of a treatment factor to the model; Odds Ratio (OR) = 0.65, 95% CI 2-sided [0.462 to 0.908] — [estimate comment as in outcome 10, analysis 1]
Statistical Analysis 2: Comparison: Durvalumab + Tremelimumab vs SoC Chemotherapy; Durvalumab + Tremelimumab Vs SoC Chemotherapy; Test type: Superiority; p = 0.093, Regression, Logistic — P-value is based on twice the change in log-likelihood resulting from the addition of a treatment factor to the model; Odds Ratio (OR) = 0.76, 95% CI 2-sided [0.543 to 1.048] — The analysis was performed using logistic regression adjusting for histology (squamous Vs non-squamous) and PD-L1 status (>=25% Vs <25%), with 95% CI calculated by profile likelihood
Statistical Analysis 3: Comparison: Durvalumab Monotherapy vs Durvalumab + Tremelimumab; Durvalumab + Tremelimumab Vs Durvalumab Monotherapy; Test type: Superiority; p = 0.406, Regression, Logistic — P-value is based on twice the change in log-likelihood resulting from the addition of a treatment factor to the model; Odds Ratio (OR) = 1.16, 95% CI 2-sided [0.818 to 1.647] — [estimate comment as in outcome 11, analysis 2]

12. Secondary Outcome: Duration of Response (DoR); PD-L1 (TC >=25%) Analysis Set Population
Description: The DoR per RECIST 1.1 using BICR assessments was defined as the time from the date of first documented response until the first date of documented progression or death in the absence of disease progression (ie, date of PFS event or censoring - date of first response + 1). The CR was defined as disappearance of all TLs (any pathological lymph nodes selected as TLs must have a reduction in short axis to <10 mm) and PR was defined as at least a 30% decrease in the sum of diameters of TLs (taking as reference the baseline sum of diameters as long as criteria for PD are not met).
Time Frame: as for outcome 2
Population: The PD-L1 (TC >=25%) analysis set included the subset of participants in the FAS whose PD-L1 status was PD-L1 (TC >=25%) as defined by the Ventana PD-L1 (SP263) assay (ie,>=25% TC expressing PD-L1 on the membrane). DoR is only analyzed for those participants with a response (including unconfirmed responses).
Measure: Median (Inter-Quartile Range); unit: months
Arm/Group | Durvalumab Monotherapy | Durvalumab + Tremelimumab | SoC Chemotherapy
Number analyzed (Participants) | 163 | 163 | 162
months | NA [4.9 to NA] — NA = Not reached. | NA [4.2 to NA] — NA = Not reached. | 4.4 [2.9 to 7.2]

13. Secondary Outcome: DoR; PD-L1 (TC >=1%) Analysis Set Population
Description: The DoR per RECIST 1.1 using BICR assessments was defined as the time from the date of first documented response (CR or PR) until the first date of documented progression or death in the absence of disease progression (ie, date of PFS event or censoring - date of first response + 1). The CR was defined as disappearance of all TLs (any pathological lymph nodes selected as TLs must have a reduction in short axis to <10 mm) and PR was defined as at least a 30% decrease in the sum of diameters of TLs (taking as reference the baseline sum of diameters as long as criteria for PD are not met).
Time Frame: as for outcome 2
Population: The PD-L1 (TC >=1%) analysis set included the subset of participants in the FAS whose PD-L1 status is PD-L1 (TC >=1%) as defined by the Ventana PD-L1 (SP263) assay (ie, >=1% TC expressing PD-L1 on the membrane). DoR is only analyzed for those participants with a response (including unconfirmed responses).
Measure: Median (Inter-Quartile Range); unit: months
Arm/Group | Durvalumab Monotherapy | Durvalumab + Tremelimumab | SoC Chemotherapy
Number analyzed (Participants) | 279 | 296 | 289
months | NA [5.5 to NA] — NA = Not reached. | NA [5.6 to NA] — NA = Not reached. | 4.4 [2.8 to 8.4]

14. Secondary Outcome: DoR; FAS Population
Description: as for outcome 12
Time Frame: as for outcome 2
Population: The FAS included all randomized participants analyzed on an ITT basis. DoR is only analyzed for those participants with a response (including unconfirmed responses).
Measure: Median (Inter-Quartile Range); unit: months
Arm/Group | Durvalumab Monotherapy | Durvalumab + Tremelimumab | SoC Chemotherapy
Number analyzed (Participants) | 374 | 372 | 372
months | NA [5.5 to NA] — NA = Not reached. | NA [4.7 to NA] — NA = Not reached. | 4.3 [2.8 to 8.4]

15. Secondary Outcome: Percentage of Participants Alive and Progression Free at 12 Months (APF12); PD-L1 (TC >=25%) Analysis Set Population
Description: The APF12 was defined as the percentage of participants who were alive and progression free per RECIST v1.1 using BICR assessments at 12 months after randomization. The PFS was calculated using the Kaplan-Meier technique.
Time Frame: Tumour scans performed at baseline then every 6 weeks up to 12 months.
Population: as for outcome 9
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Durvalumab Monotherapy | Durvalumab + Tremelimumab | SoC Chemotherapy
Number analyzed (Participants) | 163 | 163 | 162
percentage of participants | 32.3 [24.8 to 39.9] | 25.8 [18.9 to 33.1] | 14.3 [8.4 to 21.7]

16. Secondary Outcome: Percentage of Participants APF12; PD-L1 (TC >=1%) Analysis Set Population
Description: as for outcome 15
Time Frame: Tumour scans performed at baseline then every 6 weeks up to 12 months.
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Durvalumab Monotherapy | Durvalumab + Tremelimumab | SoC Chemotherapy
Number analyzed (Participants) | 279 | 296 | 289
percentage of participants | 27.0 [21.6 to 32.6] | 20.4 [15.7 to 25.5] | 14.9 [10.2 to 20.5]

17. Secondary Outcome: Percentage of Participants APF12; FAS Population
Description: as for outcome 15
Time Frame: Tumour scans performed at baseline then every 6 weeks up to 12 months.
Population: The FAS included all randomized participants analyzed on an ITT basis.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Durvalumab Monotherapy | Durvalumab + Tremelimumab | SoC Chemotherapy
Number analyzed (Participants) | 374 | 372 | 372
percentage of participants | 22.5 [18.1 to 27.1] | 19.8 [15.6 to 24.4] | 13.8 [9.7 to 18.6]

18. Secondary Outcome: Time From Randomization to Second Progression (PFS2); PD-L1 (TC >=25%) Analysis Set Population
Description: The PFS2 was defined as the time from the date of randomization to the earliest of the progression events (subsequent to that used for the primary variable PFS and excluding any confirmation of progression scans performed for first progression) or death (ie, date of PFS2 event or censoring - date of randomization + 1). The second progression event was determined by local standard clinical practice which may have included any of the following: objective radiological imaging, symptomatic progression, or death.
Time Frame: Tumour scans performed at baseline then every 6 weeks up to Week 48, then every 8 weeks thereafter until 1st progression. Disease then assessed per local practice until 2nd progression. Assessed up to data cut-off date (maximum of approximately 3 years).
Population: as for outcome 9
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Durvalumab Monotherapy | Durvalumab + Tremelimumab | SoC Chemotherapy
Number analyzed (Participants) | 163 | 163 | 162
months | 12.7 [9.4 to 16.1] | 10.9 [7.9 to 14.1] | 10.4 [9.0 to 12.5]
Statistical Analysis 1: Comparison: Durvalumab Monotherapy vs SoC Chemotherapy; Durvalumab Monotherapy Vs SoC Chemotherapy; Test type: Superiority; p = 0.030, Log Rank — [p-value comment as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.76, 95% CI 2-sided [0.597 to 0.975] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 2: Comparison: Durvalumab + Tremelimumab vs SoC Chemotherapy; Durvalumab + Tremelimumab Vs SoC Chemotherapy; Test type: Superiority; p = 0.045, Log Rank — [p-value comment as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.78, 95% CI 2-sided [0.606 to 0.994] — [estimate comment as in outcome 1, analysis 2]

19. Secondary Outcome: PFS2; PD-L1 (TC >=1%) Analysis Set Population
Description: as for outcome 18
Time Frame: as for outcome 18
Population: as for outcome 4
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Durvalumab Monotherapy | Durvalumab + Tremelimumab | SoC Chemotherapy
Number analyzed (Participants) | 279 | 296 | 289
months | 10.6 [8.0 to 12.7] | 9.4 [7.8 to 11.4] | 10.5 [9.4 to 11.7]
Statistical Analysis 1: Comparison: Durvalumab Monotherapy vs SoC Chemotherapy; Durvalumab Monotherapy Vs SoC Chemotherapy; Test type: Superiority; p = 0.255, Log Rank — [p-value comment as in outcome 4, analysis 1]; Hazard Ratio (HR) = 0.90, 95% CI 2-sided [0.746 to 1.080] — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 2: Comparison: Durvalumab + Tremelimumab vs SoC Chemotherapy; Durvalumab + Tremelimumab Vs SoC Chemotherapy; Test type: Superiority; p = 0.534, Log Rank — [p-value comment as in outcome 4, analysis 1]; Hazard Ratio (HR) = 0.94, 95% CI 2-sided [0.787 to 1.132] — [estimate comment as in outcome 4, analysis 1]

20. Secondary Outcome: PFS2; FAS Population
Description: as for outcome 18
Time Frame: as for outcome 18
Population: The FAS included all randomized participants analyzed on an ITT basis.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Durvalumab Monotherapy | Durvalumab + Tremelimumab | SoC Chemotherapy
Number analyzed (Participants) | 374 | 372 | 372
months | 9.3 [7.9 to 10.6] | 9.8 [8.8 to 11.4] | 10.1 [9.3 to 10.8]
Statistical Analysis 1: Comparison: Durvalumab Monotherapy vs SoC Chemotherapy; Durvalumab Monotherapy Vs SoC Chemotherapy; Test type: Superiority; p = 0.663, Log Rank — [p-value comment as in outcome 4, analysis 1]; Hazard Ratio (HR) = 0.97, 95% CI 2-sided [0.824 to 1.131] — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 2: Comparison: Durvalumab + Tremelimumab vs SoC Chemotherapy; Durvalumab + Tremelimumab Vs SoC Chemotherapy; Test type: Superiority; p = 0.103, Log Rank — [p-value comment as in outcome 4, analysis 1]; Hazard Ratio (HR) = 0.88, 95% CI 2-sided [0.746 to 1.027] — [estimate comment as in outcome 4, analysis 1]

21. Secondary Outcome: Change From Baseline in Disease-Related Symptoms as Assessed by European Organisation for Research and Treatment of Cancer Quality of Life Questionnaires (EORTC QLQ) at 12 Months
Description: Patient reported outcomes for 5 disease related symptoms was assessed using the EORTC QLQ-Core 30 (C30) items questionnaire (fatigue and appetite loss) and the EORTC QLQ-Lung Cancer module 13 (LC13) (dysponea, cough and chest pain). An outcome variable consisting of a score from 0 to 100 was derived for each of the symptom scales/symptom items with higher scores representing greater symptom severity. An improvement in symptoms were indicated by a negative change in score from baseline. A positive change in score from baseline indicated a deterioration of symptoms. A minimum clinically meaningful change is defined as an absolute change in the score from baseline of >=10.
Time Frame: At baseline then every 4 weeks for the first 8 weeks relative to the date of randomization, then every 8 weeks until second progression/death, whichever comes first. Assessed up to 12 months.
Population: as for outcome 9
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Durvalumab Monotherapy | Durvalumab + Tremelimumab | SoC Chemotherapy
Number analyzed (Participants) | 163 | 163 | 162
units on a scale
  EORTC QLQ-C30: Fatigue: number analyzed (Participants) | 113 | 113 | 107
  EORTC QLQ-C30: Fatigue | 1.2 (1.83) | -1.1 (1.92) | 10.6 (2.34)
  EORTC QLQ-C30: Appetite loss: number analyzed (Participants) | 113 | 113 | 107
  EORTC QLQ-C30: Appetite loss | -3.9 (2.24) | 2.4 (2.37) | 8.0 (2.83)
  EORTC QLQ-LC13: Dyspnoea: number analyzed (Participants) | 122 | 121 | 117
  EORTC QLQ-LC13: Dyspnoea | 2.3 (1.51) | 0.8 (1.60) | 5.6 (1.90)
  EORTC QLQ-LC13: Cough: number analyzed (Participants) | 122 | 121 | 117
  EORTC QLQ-LC13: Cough | -11.4 (1.88) | -5.9 (2.01) | -7.1 (2.54)
  EORTC QLQ-LC13: Chest pain: number analyzed (Participants) | 122 | 121 | 117
  EORTC QLQ-LC13: Chest pain | 0.1 (1.71) | 1.6 (1.80) | 1.7 (2.04)

22. Secondary Outcome: Serum Concentrations of Durvalumab
Description: Blood samples were collected to determine the serum concentration of durvalumab.
Time Frame: Pre-dose and within 1 hour after end of infusion at Week 0, 12 and 24, and at follow-up Month 3.
Population: Pharmacokinetic (PK) analysis set included all participants who received at least 1 dose of study treatment per the protocol for whom any post-dose data are available and who did not violate or deviate from the protocol in ways that would materially affect the PK analyses.
Measure: Mean (Standard Deviation); unit: microgram per milliliter (mcg/mL)
Arm/Group | Durvalumab Monotherapy | Durvalumab + Tremelimumab
Number analyzed (Participants) | 361 | 366
microgram per milliliter (mcg/mL)
  At Week 0: Pre-infusion: number analyzed (Participants) | 355 | 354
  At Week 0: Pre-infusion | NA (NA) — NA = Below lower limit of quantification (LLOQ). The LLOQ = 0.05 mcg/mL. | NA (NA) — NA = Below LLOQ. The LLOQ = 0.05 mcg/mL.
  At Week 0: End of infusion: number analyzed (Participants) | 353 | 349
  At Week 0: End of infusion | 484.5 (210.50) | 444.3 (150.29)
  At Week 12: Pre-infusion: number analyzed (Participants) | 185 | 187
  At Week 12: Pre-infusion | 139.5 (124.98) | 140.8 (146.25)
  At Week 12: End of infusion: number analyzed (Participants) | 177 | 179
  At Week 12: End of infusion | 625.3 (453.8) | 506.1 (231.89)
  At Week 24: Pre-infusion: number analyzed (Participants) | 136 | 123
  At Week 24: Pre-infusion | 163.0 (170.04) | 197.0 (228.79)
  At Week 24: End of infusion: number analyzed (Participants) | 135 | 123
  At Week 24: End of infusion | 598.2 (344.52) | 553.2 (193.33)
  At follow-up Month 3: number analyzed (Participants) | 42 | 32
  At follow-up Month 3 | 49.3 (132.54) | 41.4 (131.71)

23. Secondary Outcome: Serum Concentrations of Tremelimumab
Description: Blood samples were collected to determine the serum concentration of tremelimumab.
Time Frame: Pre-dose and within 1 hour after end of infusion at Week 0 and 12, and at follow-up Month 3.
Population: The PK analysis set included all participants who received at least 1 dose of study treatment per the protocol for whom any post-dose data are available and who did not violate or deviate from the protocol in ways that would materially affect the PK analyses.
Measure: Mean (Standard Deviation); unit: mcg/mL
Arm/Group | Durvalumab + Tremelimumab
Number analyzed (Participants) | 366
mcg/mL
  At Week 0: Pre-infusion: number analyzed (Participants) | 358
  At Week 0: Pre-infusion | NA (NA) — NA = Below LLOQ. The LLOQ = 0.05 mcg/mL.
  At Week 0: End of infusion: number analyzed (Participants) | 359
  At Week 0: End of infusion | 22.6 (14.84)
  At Week 12: Pre-infusion: number analyzed (Participants) | 187
  At Week 12: Pre-infusion | 4.9 (4.16)
  At Week 12: End of infusion: number analyzed (Participants) | 180
  At Week 12: End of infusion | 24.8 (10.43)
  At follow-up Month 3: number analyzed (Participants) | 28
  At follow-up Month 3 | 0.5 (0.42)

24. Secondary Outcome: Maximum Serum Concentration at Steady State (Cmax_ss) of Durvalumab
Description: Blood samples were collected to determine the Cmax_ss of durvalumab. Steady state was defined as Cycle 4 (Week 12). PK parameters were determined using standard non-compartmental methods.
Time Frame: Within 1 hour after end of infusion on infusion day at Week 12.
Population: as for outcome 23
Measure: Mean (Standard Deviation); unit: mcg/mL
Arm/Group | Durvalumab Monotherapy | Durvalumab + Tremelimumab
Number analyzed (Participants) | 361 | 366
mcg/mL | 625.3 (453.80) | 506.1 (231.89)

25. Secondary Outcome: Cmax_ss of Tremelimumab
Description: Blood samples were collected to determine the Cmax_ss of tremelimumab. Steady state was defined as Cycle 4 (Week 12). PK parameters were determined using standard non-compartmental methods.
Time Frame: Within 1 hour after end of infusion on infusion day at Week 12.
Population: as for outcome 23
Measure: Mean (Standard Deviation); unit: mcg/mL
Arm/Group | Durvalumab + Tremelimumab
Number analyzed (Participants) | 366
mcg/mL | 24.8 (10.43)

26. Secondary Outcome: Trough Serum Concentration at Steady State (Ctrough_ss) of Durvalumab
Description: Blood samples were collected to determine the Ctrough_ss of durvalumab. Steady state was defined as Cycle 4 (Week 12). PK parameters were determined using standard non-compartmental methods.
Time Frame: Pre-dose at Week 12.
Population: as for outcome 23
Measure: Mean (Standard Deviation); unit: mcg/mL
Arm/Group | Durvalumab Monotherapy | Durvalumab + Tremelimumab
Number analyzed (Participants) | 361 | 366
mcg/mL | 139.5 (124.98) | 140.8 (146.25)

27. Secondary Outcome: Ctrough_ss of Tremelimumab
Description: Blood samples were collected to determine the Ctrough_ss of tremelimumab. Steady state was defined as Cycle 4 (Week 12). PK parameters were determined using standard non-compartmental methods.
Time Frame: Pre-dose at Week 12.
Population: as for outcome 23
Measure: Mean (Standard Deviation); unit: mcg/mL
Arm/Group | Durvalumab + Tremelimumab
Number analyzed (Participants) | 366
mcg/mL | 4.9 (4.16)

28. Secondary Outcome: Number of Participants With Anti-Drug Antibody (ADA) Response to Durvalumab
Description: Blood samples were measured for the presence of ADAs and ADA-neutralizing antibodies (nAb) for durvalumab using validated assays. Tiered analysis was performed to include screening, confirmatory, and titer assay components, and positive-negative cut points previously statistically determined from drug-naïve validation samples were employed. Immunogenicity results were analyzed by summarizing the number of participants who developed detectable ADAs against durvalumab. Persistently positive is defined as having at least 2 post-baseline ADA positive measurements with at least 16 weeks (112 days) between the first and last positive measurements, or an ADA positive result at the last available assessment. Transiently positive is defined as having at least one post-baseline ADA positive measurement and not fulfilling the conditions for persistently positive.
Time Frame: At Weeks 0, 12, and 24; 3 and 6 months after last dose of study treatment.
Population: Safety analysis set included all participants who received at least 1 dose of study treatment. ADA evaluable population included participants who have non-missing durvalumab baseline ADA and at least one non-missing post-baseline durvalumab ADA result.
Measure: Count of Participants; unit: Participants
Arm/Group | Durvalumab Monotherapy | Durvalumab + Tremelimumab
Number analyzed (Participants) | 212 | 223
Participants
  ADA positive at any time | 17 | 14
  Treatment-emergent ADA positive | 8 | 8
  ADA positive at baseline and post-baseline | 3 | 1
  ADA positive at post-baseline only | 8 | 8
  ADA positive at baseline only | 6 | 5
  Treatment-boosted ADA | 0 | 0
  Persistent positive | 8 | 9
  Transient positive | 3 | 0
  nAb positive at any visit | 2 | 1

29. Secondary Outcome: Number of Participants With ADA Response to Tremelimumab
Description: Blood samples were measured for the presence of ADAs and ADA-nAb for tremelimumab using validated assays. Tiered analysis was performed to include screening, confirmatory, and titer assay components, and positive-negative cut points previously statistically determined from drug-naïve validation samples were employed. Immunogenicity results were analyzed by summarizing the number of participants who developed detectable ADAs against tremelimumab. Persistently positive is defined as having at least 2 post-baseline ADA positive measurements with at least 16 weeks (112 days) between the first and last positive measurements, or an ADA positive result at the last available assessment. Transiently positive is defined as having at least one post-baseline ADA positive measurement and not fulfilling the conditions for persistently positive.
Time Frame: At Weeks 0 and 12; 3 and 6 months after last dose of study treatment.
Population: Safety analysis set included all participants who received at least 1 dose of study treatment. ADA evaluable population included participants who have non-missing baseline tremelimumab ADA and at least one non-missing post-baseline tremelimumab ADA result.
Measure: Count of Participants; unit: Participants
Arm/Group | Durvalumab + Tremelimumab
Number analyzed (Participants) | 219
Participants
  ADA positive at any time | 33
  Treatment-emergent ADA positive | 28
  ADA positive at baseline and post-baseline | 1
  ADA positive at post-baseline only | 28
  ADA positive at baseline only | 4
  Treatment-boosted ADA | 0
  Persistent positive | 25
  Transient positive | 4
  nAb positive at any visit | 25

ADVERSE EVENTS:
Time Frame: From first administration of study treatment up to 90 days after last dose of durvalumab and tremelimumab or 30 days after last dose of SoC or date of initiation of the first subsequent therapy, whichever occurs first, approximately 3 years. All-cause mortality, from screening up to data cut-off date (approximately 3 years 1 month).
Description: Safety analysis set included all participants who received at least 1 dose of study treatment. All-cause mortality was determined for participants in FAS.
Arm/Group | Durvalumab Monotherapy | Durvalumab + Tremelimumab | SoC Chemotherapy
All-Cause Mortality (participants affected / at risk) | 278/374 | 278/372 | 297/372
Serious Adverse Events (participants affected / at risk) | 131/369 | 178/371 | 112/352
Other Adverse Events (participants affected / at risk) | 335/369 | 328/371 | 332/352
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Durvalumab Monotherapy (N=369) | Durvalumab + Tremelimumab (N=371) | SoC Chemotherapy (N=352)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 4 (5) | 14 (18)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 2 (2)
Immune thrombocytopenic purpura (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Pancytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 6 (6)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 2 (2)
Acute coronary syndrome (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 2 (3) | 5 (5) | 1 (1)
Atrial flutter (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Bradycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Cardiac arrest (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Cardiac failure (Cardiac disorders) | 1 (1) | 3 (3) | 0 (0)
Cardiac tamponade (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0)
Myocardial ischaemia (Cardiac disorders) | 0 (0) | 2 (3) | 0 (0)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Pericardial effusion (Cardiac disorders) | 3 (3) | 0 (0) | 0 (0)
Pericarditis (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Wolff-Parkinson-White syndrome (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Adrenal insufficiency (Endocrine disorders) | 1 (1) | 2 (2) | 0 (0)
Autoimmune thyroiditis (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0)
Hypophysitis (Endocrine disorders) | 0 (0) | 2 (2) | 0 (0)
Hypothyroidism (Endocrine disorders) | 3 (3) | 0 (0) | 0 (0)
Secondary adrenocortical insufficiency (Endocrine disorders) | 0 (0) | 2 (2) | 0 (0)
Secondary hypothyroidism (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0)
Vitreous haemorrhage (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (2)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Autoimmune colitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Cheilitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 2 (2) | 6 (6) | 0 (0)
Colitis ischaemic (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Colitis microscopic (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 2 (2) | 2 (2) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 12 (15) | 6 (7)
Dysphagia (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0)
Enterocolitis (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Faecaloma (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Gastric haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastric perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Gastrointestinal disorder (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Impaired gastric emptying (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Intestinal ischaemia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Melaena (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (2) | 3 (4)
Oesophageal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Oesophagitis (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Peptic ulcer haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Rectal ulcer haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Small intestinal perforation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 4 (4) | 1 (2) | 2 (2)
Asthenia (General disorders) | 0 (0) | 2 (2) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1)
Death (General disorders) | 1 (1) | 1 (1) | 1 (1)
Euthanasia (General disorders) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 0 (0) | 6 (6) | 0 (0)
Feeling abnormal (General disorders) | 1 (1) | 0 (0) | 0 (0)
General physical health deterioration (General disorders) | 1 (1) | 3 (3) | 2 (3)
Generalised oedema (General disorders) | 1 (1) | 1 (1) | 1 (1)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 1 (1)
Malaise (General disorders) | 0 (0) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1) | 1 (1)
Oedema peripheral (General disorders) | 1 (1) | 0 (0) | 2 (2)
Pyrexia (General disorders) | 5 (5) | 4 (4) | 1 (1)
Sudden death (General disorders) | 1 (1) | 2 (2) | 0 (0)
Acute hepatic failure (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Bile duct obstruction (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Bile duct stenosis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Cholangitis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Drug-induced liver injury (Hepatobiliary disorders) | 1 (1) | 5 (5) | 0 (0)
Hepatitis (Hepatobiliary disorders) | 1 (1) | 2 (2) | 0 (0)
Hepatitis acute (Hepatobiliary disorders) | 1 (1) | 1 (1) | 0 (0)
Hepatotoxicity (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Anaphylactic reaction (Immune system disorders) | 2 (2) | 0 (0) | 0 (0)
Anaphylactic shock (Immune system disorders) | 0 (0) | 1 (1) | 1 (1)
Drug hypersensitivity (Immune system disorders) | 1 (1) | 1 (1) | 1 (2)
Abdominal abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Arthritis bacterial (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 3 (3)
Clostridium difficile colitis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Device related infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Empyema (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Erysipelas (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Febrile infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Herpes zoster (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Infective spondylitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 2 (2) | 0 (0) | 1 (1)
Lung infection (Infections and infestations) | 2 (2) | 1 (2) | 3 (3)
Pleural infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pneumocystis jirovecii pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 20 (27) | 21 (28) | 19 (22)
Pneumonia bacterial (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Pneumonia cytomegaloviral (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pneumonia legionella (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pneumonia staphylococcal (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pneumonia streptococcal (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Post procedural infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Postoperative wound infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pulmonary sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Puncture site infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 5 (5)
Respiratory tract infection bacterial (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 3 (3) | 3 (3) | 2 (2)
Septic shock (Infections and infestations) | 3 (3) | 2 (2) | 1 (1)
Skin infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Soft tissue infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 1 (1) | 3 (3)
Urosepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Wound infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Pneumocephalus (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Procedural pneumothorax (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Radiation pneumonitis (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0)
Spinal fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Subdural haemorrhage (Injury, poisoning and procedural complications) | 1 (2) | 0 (0) | 0 (0)
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Traumatic fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Upper limb fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Wound complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Wound secretion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Blood calcium increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 1 (1) | 1 (1) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
C-reactive protein increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Haemoglobin decreased (Investigations) | 0 (0) | 1 (1) | 1 (1)
Lipase increased (Investigations) | 1 (1) | 3 (3) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 2 (2)
Troponin increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 5 (6) | 1 (1)
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Fulminant type 1 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (2)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 3 (3) | 1 (1)
Hypophagia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2)
Malnutrition (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Vitamin B1 deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Groin pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Polyarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Rectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Altered state of consciousness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Basal ganglia infarction (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Basilar artery stenosis (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Cerebral infarction (Nervous system disorders) | 2 (2) | 2 (2) | 0 (0)
Cerebral ischaemia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1)
Depressed level of consciousness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Epilepsy (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0)
Facial neuralgia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Generalised tonic-clonic seizure (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Hydrocephalus (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Hypoglycaemic coma (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 2 (3) | 1 (1) | 0 (0)
Lethargy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Monoplegia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Neurotoxicity (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Paraplegia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Sciatica (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 2 (5) | 0 (0)
Sensory loss (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 2 (2) | 2 (2) | 1 (1)
Alcohol withdrawal syndrome (Psychiatric disorders) | 0 (0) | 1 (3) | 0 (0)
Completed suicide (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Confusional state (Psychiatric disorders) | 4 (4) | 1 (1) | 0 (0)
Delirium (Psychiatric disorders) | 1 (2) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 2 (2) | 0 (0)
Logorrhoea (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Mental status changes (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Organic brain syndrome (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1)
Azotaemia (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Nephritis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 2 (2)
Renal infarct (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0)
Prostatitis (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 1 (1)
Alveolitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2 (4) | 7 (7) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 6 (7) | 2 (2)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Emphysema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (2) | 4 (4)
Hypercapnia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 7 (8) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 5 (5) | 1 (1)
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 9 (9) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 2 (2) | 0 (0)
Pneumothorax spontaneous (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 6 (6) | 8 (8)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 1 (1)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Diabetic foot (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Pemphigoid (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Toxic skin eruption (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Blood pressure inadequately controlled (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 2 (2) | 0 (0)
Embolism (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Peripheral artery occlusion (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Peripheral embolism (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Peripheral ischaemia (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Superior vena cava syndrome (Vascular disorders) | 1 (1) | 2 (2) | 0 (0)
Thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Vasoconstriction (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Durvalumab Monotherapy (N=369) | Durvalumab + Tremelimumab (N=371) | SoC Chemotherapy (N=352)
Anaemia (Blood and lymphatic system disorders) | 36 (37) | 33 (39) | 136 (177)
Bone marrow failure (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (2)
Coagulopathy (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Cytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Eosinophilia (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 2 (2)
Granulocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Hypercoagulation (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 8 (8) | 4 (4) | 3 (3)
Leukopenia (Blood and lymphatic system disorders) | 2 (2) | 1 (1) | 15 (32)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (1) | 2 (2) | 0 (0)
Lymphopenia (Blood and lymphatic system disorders) | 3 (3) | 2 (2) | 2 (3)
Neutropenia (Blood and lymphatic system disorders) | 6 (8) | 2 (2) | 65 (123)
Neutrophilia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Pancytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 3 (4)
Spontaneous haematoma (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 3 (3) | 8 (9) | 45 (68)
Thrombocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 2 (2)
Acute left ventricular failure (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Angina pectoris (Cardiac disorders) | 2 (2) | 1 (2) | 1 (1)
Arrhythmia (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0)
Arteriosclerosis coronary artery (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 6 (6) | 3 (3) | 6 (7)
Bradycardia (Cardiac disorders) | 0 (0) | 2 (2) | 1 (1)
Cardiac arrest (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
Cardiac failure (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Cardiac flutter (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Cardiomegaly (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Diastolic dysfunction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Hepatojugular reflux (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Left atrial enlargement (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Myocardial ischaemia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Palpitations (Cardiac disorders) | 2 (2) | 3 (3) | 1 (1)
Pericardial effusion (Cardiac disorders) | 0 (0) | 2 (2) | 2 (2)
Pericarditis (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 3 (3) | 0 (0)
Stress cardiomyopathy (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Supraventricular extrasystoles (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 1 (1) | 3 (3) | 1 (1)
Tachyarrhythmia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 5 (5) | 5 (5) | 5 (5)
Tricuspid valve incompetence (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Cerumen impaction (Ear and labyrinth disorders) | 2 (2) | 0 (0) | 0 (0)
Deafness (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 1 (1)
Deafness unilateral (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Ear discomfort (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 1 (1) | 2 (2) | 2 (2)
Ear pruritus (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Excessive cerumen production (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Hypoacusis (Ear and labyrinth disorders) | 0 (0) | 6 (6) | 2 (2)
Otorrhoea (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Ototoxicity (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 2 (2)
Tinnitus (Ear and labyrinth disorders) | 2 (2) | 3 (4) | 12 (12)
Vertigo (Ear and labyrinth disorders) | 2 (2) | 6 (7) | 5 (5)
Vertigo positional (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1)
Adrenal insufficiency (Endocrine disorders) | 1 (1) | 6 (6) | 1 (1)
Autoimmune thyroiditis (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1)
Cushingoid (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1)
Euthyroid sick syndrome (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 12 (12) | 24 (25) | 2 (2)
Hypothyroidism (Endocrine disorders) | 26 (28) | 32 (34) | 2 (2)
Primary hypothyroidism (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0)
Thyroid mass (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0)
Thyroiditis (Endocrine disorders) | 2 (2) | 2 (2) | 0 (0)
Age-related macular degeneration (Eye disorders) | 0 (0) | 1 (2) | 0 (0)
Angle closure glaucoma (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Blepharitis (Eye disorders) | 0 (0) | 1 (1) | 1 (1)
Blindness (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Blindness transient (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Cataract (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Conjunctival haemorrhage (Eye disorders) | 1 (1) | 0 (0) | 1 (1)
Conjunctivitis allergic (Eye disorders) | 0 (0) | 1 (1) | 1 (1)
Diplopia (Eye disorders) | 4 (4) | 3 (4) | 0 (0)
Dry eye (Eye disorders) | 12 (13) | 4 (4) | 9 (9)
Episcleritis (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Extraocular muscle paresis (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Eye haemorrhage (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Eye irritation (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Eye pain (Eye disorders) | 1 (1) | 1 (1) | 0 (0)
Eye pruritus (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Eye swelling (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Eye ulcer (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Eyelid oedema (Eye disorders) | 0 (0) | 0 (0) | 2 (2)
Eyelid ptosis (Eye disorders) | 1 (1) | 2 (2) | 0 (0)
Glaucoma (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Halo vision (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Keratitis (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Lacrimation increased (Eye disorders) | 3 (3) | 2 (2) | 15 (15)
Neovascular age-related macular degeneration (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Ocular hyperaemia (Eye disorders) | 1 (1) | 1 (1) | 0 (0)
Ocular hypertension (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Periorbital oedema (Eye disorders) | 1 (1) | 1 (1) | 0 (0)
Photopsia (Eye disorders) | 0 (0) | 1 (1) | 1 (1)
Polypoidal choroidal vasculopathy (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Pterygium (Eye disorders) | 0 (0) | 0 (0) | 1 (2)
Punctate keratitis (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Uveitis (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Vision blurred (Eye disorders) | 5 (5) | 5 (5) | 5 (5)
Visual acuity reduced (Eye disorders) | 1 (1) | 1 (1) | 2 (2)
Visual impairment (Eye disorders) | 1 (1) | 3 (3) | 1 (1)
Vitreous floaters (Eye disorders) | 2 (2) | 1 (2) | 0 (0)
Xerophthalmia (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 2 (2) | 4 (4) | 2 (2)
Abdominal distension (Gastrointestinal disorders) | 4 (5) | 4 (5) | 5 (5)
Abdominal pain (Gastrointestinal disorders) | 15 (16) | 17 (18) | 7 (8)
Abdominal pain lower (Gastrointestinal disorders) | 1 (1) | 0 (0) | 3 (3)
Abdominal pain upper (Gastrointestinal disorders) | 13 (14) | 9 (9) | 15 (15)
Abdominal tenderness (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Abnormal faeces (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Anal fistula (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Anal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Anal incontinence (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Anal pruritus (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Anorectal discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Aphthous ulcer (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Ascites (Gastrointestinal disorders) | 1 (1) | 2 (2) | 1 (1)
Cheilitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Chilaiditi's syndrome (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Chronic gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (2)
Colitis (Gastrointestinal disorders) | 1 (1) | 6 (7) | 0 (0)
Colitis ulcerative (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 62 (69) | 59 (67) | 83 (99)
Crohn's disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Dental caries (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 51 (71) | 74 (117) | 41 (58)
Diarrhoea haemorrhagic (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 8 (8) | 19 (20) | 4 (4)
Duodenal ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Duodenitis (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 13 (13) | 11 (12) | 19 (20)
Dysphagia (Gastrointestinal disorders) | 11 (12) | 10 (11) | 6 (6)
Enterocolitis (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Epigastric discomfort (Gastrointestinal disorders) | 0 (0) | 2 (3) | 4 (4)
Eructation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Faecaloma (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Faeces discoloured (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (2)
Faeces soft (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 5 (5) | 3 (3)
Food poisoning (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Frequent bowel movements (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Gastric ulcer (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1)
Gastritis (Gastrointestinal disorders) | 2 (2) | 6 (6) | 2 (3)
Gastritis erosive (Gastrointestinal disorders) | 0 (0) | 3 (3) | 0 (0)
Gastritis haemorrhagic (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 6 (7) | 7 (8) | 8 (8)
Gingival swelling (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Glossodynia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Haemorrhagic erosive gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1 (1) | 2 (2) | 1 (1)
Haemorrhoids (Gastrointestinal disorders) | 1 (1) | 1 (1) | 4 (4)
Hiatus hernia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Hypoaesthesia oral (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Ileus (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Large intestine polyp (Gastrointestinal disorders) | 1 (1) | 2 (2) | 1 (1)
Lip swelling (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Lip ulceration (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Melaena (Gastrointestinal disorders) | 2 (2) | 3 (3) | 2 (2)
Mouth haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2)
Mouth swelling (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Mouth ulceration (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1)
Nausea (Gastrointestinal disorders) | 46 (53) | 78 (96) | 143 (215)
Odynophagia (Gastrointestinal disorders) | 3 (3) | 1 (1) | 1 (1)
Oesophageal stenosis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Oesophagitis (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Oral discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Oral dysaesthesia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Oral mucosal blistering (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Oral mucosal erythema (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Oral pain (Gastrointestinal disorders) | 2 (3) | 2 (2) | 2 (2)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Paraesthesia oral (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Peptic ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Peritoneal disorder (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Proctalgia (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Rectal tenesmus (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Rectal ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Salivary hypersecretion (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 9 (9) | 13 (15) | 29 (41)
Subileus (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Tongue discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Tongue ulceration (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 5 (5) | 2 (2) | 2 (2)
Umbilical hernia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 28 (32) | 30 (35) | 74 (93)
Asthenia (General disorders) | 48 (63) | 45 (50) | 48 (70)
Axillary pain (General disorders) | 1 (1) | 0 (0) | 1 (1)
Catheter site bruise (General disorders) | 1 (1) | 0 (0) | 0 (0)
Catheter site erosion (General disorders) | 1 (1) | 0 (0) | 0 (0)
Catheter site erythema (General disorders) | 0 (0) | 0 (0) | 1 (1)
Catheter site inflammation (General disorders) | 1 (1) | 0 (0) | 0 (0)
Catheter site pain (General disorders) | 2 (2) | 2 (2) | 2 (2)
Chest discomfort (General disorders) | 0 (0) | 0 (0) | 1 (1)
Chest pain (General disorders) | 5 (5) | 2 (2) | 1 (1)
Chills (General disorders) | 7 (7) | 10 (12) | 8 (9)
Extravasation (General disorders) | 0 (0) | 0 (0) | 1 (1)
Face oedema (General disorders) | 2 (2) | 0 (0) | 2 (2)
Facial pain (General disorders) | 3 (3) | 0 (0) | 1 (1)
Fatigue (General disorders) | 65 (72) | 80 (95) | 80 (92)
Feeling abnormal (General disorders) | 1 (1) | 0 (0) | 0 (0)
Feeling cold (General disorders) | 2 (3) | 1 (1) | 0 (0)
Feeling hot (General disorders) | 0 (0) | 0 (0) | 1 (1)
Gait disturbance (General disorders) | 1 (1) | 1 (1) | 1 (2)
General physical health deterioration (General disorders) | 3 (3) | 2 (2) | 2 (2)
Generalised oedema (General disorders) | 1 (1) | 1 (1) | 0 (0)
Hyperthermia (General disorders) | 0 (0) | 1 (1) | 1 (3)
Impaired healing (General disorders) | 1 (1) | 0 (0) | 0 (0)
Inflammation (General disorders) | 1 (1) | 0 (0) | 2 (2)
Influenza like illness (General disorders) | 7 (8) | 8 (10) | 4 (5)
Infusion site extravasation (General disorders) | 0 (0) | 1 (1) | 1 (1)
Injection site bruising (General disorders) | 0 (0) | 0 (0) | 1 (1)
Injection site erythema (General disorders) | 1 (1) | 0 (0) | 0 (0)
Injection site swelling (General disorders) | 1 (1) | 0 (0) | 4 (4)
Localised oedema (General disorders) | 1 (1) | 0 (0) | 1 (1)
Malaise (General disorders) | 9 (9) | 7 (11) | 8 (8)
Mass (General disorders) | 0 (0) | 1 (1) | 0 (0)
Medical device site inflammation (General disorders) | 1 (1) | 0 (0) | 0 (0)
Mucosal dryness (General disorders) | 0 (0) | 1 (1) | 0 (0)
Mucosal inflammation (General disorders) | 1 (1) | 1 (1) | 2 (2)
Mucosal membrane hyperplasia (General disorders) | 1 (1) | 0 (0) | 0 (0)
Mucous membrane disorder (General disorders) | 0 (0) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 9 (9) | 10 (11) | 9 (9)
Oedema (General disorders) | 6 (7) | 4 (4) | 12 (15)
Oedema peripheral (General disorders) | 30 (39) | 29 (32) | 28 (33)
Pain (General disorders) | 4 (4) | 7 (7) | 3 (3)
Performance status decreased (General disorders) | 0 (0) | 0 (0) | 1 (1)
Peripheral swelling (General disorders) | 5 (5) | 2 (2) | 4 (4)
Polyp (General disorders) | 0 (0) | 1 (1) | 0 (0)
Puncture site pain (General disorders) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 36 (46) | 39 (47) | 25 (36)
Stenosis (General disorders) | 0 (0) | 1 (1) | 0 (0)
Swelling (General disorders) | 1 (1) | 0 (0) | 1 (1)
Tenderness (General disorders) | 0 (0) | 1 (1) | 0 (0)
Vaccination site oedema (General disorders) | 0 (0) | 0 (0) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Cholestasis (Hepatobiliary disorders) | 1 (1) | 2 (2) | 2 (2)
Hepatic congestion (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Hepatic cyst (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Hepatic function abnormal (Hepatobiliary disorders) | 3 (3) | 4 (6) | 1 (1)
Hepatic steatosis (Hepatobiliary disorders) | 0 (0) | 2 (2) | 0 (0)
Hepatitis (Hepatobiliary disorders) | 0 (0) | 2 (2) | 0 (0)
Hepatitis toxic (Hepatobiliary disorders) | 1 (1) | 0 (0) | 1 (1)
Hepatocellular injury (Hepatobiliary disorders) | 0 (0) | 1 (1) | 1 (1)
Hepatotoxicity (Hepatobiliary disorders) | 0 (0) | 0 (0) | 2 (2)
Immune-mediated hepatitis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Allergic oedema (Immune system disorders) | 0 (0) | 1 (1) | 0 (0)
Allergy to fermented products (Immune system disorders) | 0 (0) | 1 (1) | 0 (0)
Anaphylactic reaction (Immune system disorders) | 1 (1) | 0 (0) | 0 (0)
Contrast media allergy (Immune system disorders) | 2 (2) | 5 (6) | 1 (1)
Contrast media reaction (Immune system disorders) | 0 (0) | 2 (2) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 4 (4) | 1 (1) | 1 (1)
Food allergy (Immune system disorders) | 1 (1) | 0 (0) | 0 (0)
Hypersensitivity (Immune system disorders) | 1 (1) | 3 (3) | 0 (0)
Seasonal allergy (Immune system disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Abscess oral (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Aspergillus infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Biliary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Bronchiolitis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Bronchitis (Infections and infestations) | 10 (11) | 14 (15) | 10 (10)
Bronchitis viral (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Candida infection (Infections and infestations) | 1 (1) | 3 (3) | 2 (2)
Carbuncle (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 2 (2) | 2 (2)
Chest wall abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Clostridium colitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Conjunctivitis (Infections and infestations) | 5 (5) | 7 (9) | 13 (14)
Cystitis (Infections and infestations) | 3 (3) | 2 (2) | 1 (1)
Cytomegalovirus infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Device related infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Ear infection (Infections and infestations) | 1 (1) | 2 (2) | 0 (0)
Endocarditis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Epididymitis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Erysipelas (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Eyelid infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Folliculitis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Fungal pharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Fungal skin infection (Infections and infestations) | 3 (3) | 2 (2) | 0 (0)
Gangrene (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 3 (3) | 2 (2) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Gingivitis (Infections and infestations) | 1 (1) | 1 (1) | 1 (1)
Groin abscess (Infections and infestations) | 1 (2) | 0 (0) | 0 (0)
Helicobacter infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Herpes simplex (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Herpes zoster (Infections and infestations) | 2 (2) | 7 (7) | 4 (4)
Herpes zoster oticus (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Hordeolum (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Impetigo (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Infected dermal cyst (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Infection (Infections and infestations) | 2 (2) | 3 (3) | 2 (2)
Influenza (Infections and infestations) | 8 (8) | 5 (6) | 4 (5)
Intervertebral discitis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Lip infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Localised infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Lower respiratory tract infection (Infections and infestations) | 5 (7) | 2 (3) | 1 (1)
Lung infection (Infections and infestations) | 4 (4) | 6 (7) | 3 (4)
Lung infection pseudomonal (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Medical device site infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Mucosal infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (2)
Nasopharyngitis (Infections and infestations) | 13 (19) | 16 (27) | 16 (18)
Oral candidiasis (Infections and infestations) | 2 (2) | 6 (6) | 4 (5)
Oral fungal infection (Infections and infestations) | 2 (2) | 1 (1) | 0 (0)
Oral herpes (Infections and infestations) | 2 (2) | 0 (0) | 3 (3)
Oral infection (Infections and infestations) | 1 (1) | 1 (1) | 1 (1)
Otitis media (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Parainfluenzae virus infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Paronychia (Infections and infestations) | 2 (2) | 2 (2) | 0 (0)
Pelvic infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Periodontitis (Infections and infestations) | 1 (1) | 0 (0) | 2 (2)
Perirectal abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pharyngitis (Infections and infestations) | 3 (3) | 3 (3) | 2 (2)
Pneumonia (Infections and infestations) | 16 (19) | 13 (14) | 7 (7)
Pneumonia bacterial (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pneumonia necrotising (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Post procedural infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Postoperative wound infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pseudomembranous colitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pulmonary tuberculosis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pulpitis dental (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pyelonephritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pyoderma (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pyuria (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Rash pustular (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Respiratory tract infection (Infections and infestations) | 12 (14) | 6 (6) | 7 (9)
Respiratory tract infection viral (Infections and infestations) | 2 (2) | 3 (4) | 3 (5)
Rhinitis (Infections and infestations) | 5 (7) | 3 (3) | 4 (4)
Sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Severe acute respiratory syndrome (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Sialoadenitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 6 (8) | 7 (9) | 3 (3)
Skin infection (Infections and infestations) | 2 (2) | 1 (1) | 1 (1)
Soft tissue infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (2)
Staphylococcal infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Subcutaneous abscess (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Sweating fever (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Tinea versicolour (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Tooth abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Tooth infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Tracheobronchitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 18 (23) | 12 (19) | 11 (12)
Urinary tract infection (Infections and infestations) | 12 (14) | 8 (11) | 9 (11)
Vestibular neuronitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Viral infection (Infections and infestations) | 1 (1) | 2 (2) | 0 (0)
Vulvovaginal candidiasis (Infections and infestations) | 1 (2) | 0 (0) | 0 (0)
Vulvovaginal mycotic infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Wound infection (Infections and infestations) | 2 (2) | 1 (1) | 0 (0)
Acetabulum fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Animal bite (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Arthropod sting (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Bone fissure (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Chest injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1)
Clavicle fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 3 (4) | 3 (3) | 2 (2)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 4 (8) | 4 (4)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Foreign body in gastrointestinal tract (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Fractured sacrum (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Hand fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 4 (4) | 2 (2) | 0 (0)
Joint injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Laceration (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Muscle strain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Neck injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Palate injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Post procedural fever (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Post procedural haematuria (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Post-traumatic pain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Postoperative wound complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1) | 2 (2) | 3 (3)
Procedural pneumothorax (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Radiation injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Radiation oesophagitis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Radiation pneumonitis (Injury, poisoning and procedural complications) | 3 (3) | 0 (0) | 0 (0)
Radiation skin injury (Injury, poisoning and procedural complications) | 3 (3) | 1 (1) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 2 (3) | 1 (1) | 0 (0)
Skeletal injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Skin abrasion (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 1 (1)
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Toxicity to various agents (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Transfusion reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Traumatic intracranial haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Upper limb fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Vascular access complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Wound (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0)
Wound complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (3) | 0 (0)
Activated partial thromboplastin time prolonged (Investigations) | 0 (0) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 17 (19) | 22 (24) | 18 (21)
Amylase increased (Investigations) | 15 (17) | 18 (23) | 6 (6)
Aspartate aminotransferase increased (Investigations) | 13 (14) | 22 (24) | 14 (16)
Blood albumin increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Blood alkaline phosphatase decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 12 (13) | 18 (22) | 7 (7)
Blood bilirubin increased (Investigations) | 2 (4) | 7 (7) | 4 (5)
Blood calcium decreased (Investigations) | 1 (1) | 1 (1) | 0 (0)
Blood cholesterol increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Blood creatine phosphokinase increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 5 (6) | 15 (20) | 18 (22)
Blood electrolytes increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Blood glucose increased (Investigations) | 2 (5) | 1 (1) | 1 (1)
Blood lactate dehydrogenase abnormal (Investigations) | 0 (0) | 0 (0) | 1 (1)
Blood lactate dehydrogenase increased (Investigations) | 5 (7) | 4 (5) | 5 (5)
Blood lactic acid increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Blood magnesium increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Blood pressure increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Blood sodium decreased (Investigations) | 1 (1) | 1 (1) | 0 (0)
Blood thyroid stimulating hormone decreased (Investigations) | 1 (1) | 4 (4) | 0 (0)
Blood thyroid stimulating hormone increased (Investigations) | 3 (4) | 4 (4) | 0 (0)
Blood urea increased (Investigations) | 1 (1) | 1 (1) | 2 (2)
Blood uric acid decreased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Blood uric acid increased (Investigations) | 2 (2) | 1 (1) | 1 (1)
Body temperature increased (Investigations) | 0 (0) | 2 (3) | 1 (2)
Brain natriuretic peptide increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
C-reactive protein increased (Investigations) | 4 (4) | 4 (6) | 8 (10)
Carbon dioxide decreased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Computerised tomogram thorax abnormal (Investigations) | 1 (1) | 0 (0) | 0 (0)
Cortisol decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Creatinine renal clearance decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Ejection fraction decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Fibrin D dimer increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Gamma-glutamyltransferase increased (Investigations) | 13 (19) | 12 (13) | 12 (12)
Haematocrit decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Haemoglobin decreased (Investigations) | 1 (1) | 0 (0) | 1 (2)
Haemoglobin increased (Investigations) | 1 (1) | 1 (1) | 0 (0)
Hepatic enzyme increased (Investigations) | 1 (1) | 0 (0) | 2 (2)
International normalised ratio increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Intraocular pressure increased (Investigations) | 1 (1) | 1 (1) | 0 (0)
Lipase increased (Investigations) | 8 (9) | 15 (22) | 6 (8)
Liver function test abnormal (Investigations) | 0 (0) | 1 (1) | 0 (0)
Liver function test decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Liver function test increased (Investigations) | 3 (3) | 1 (1) | 2 (2)
Lymph node palpable (Investigations) | 0 (0) | 1 (1) | 0 (0)
Lymphocyte count decreased (Investigations) | 4 (6) | 4 (6) | 7 (10)
Monocyte count decreased (Investigations) | 0 (0) | 2 (2) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 1 (1) | 23 (52)
Platelet count decreased (Investigations) | 3 (3) | 4 (4) | 20 (34)
Platelet count increased (Investigations) | 1 (1) | 0 (0) | 1 (1)
Protein total decreased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Protein urine present (Investigations) | 1 (1) | 1 (1) | 0 (0)
Prothrombin time prolonged (Investigations) | 0 (0) | 0 (0) | 1 (1)
Red blood cell count decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Red blood cells urine (Investigations) | 1 (1) | 0 (0) | 0 (0)
Staphylococcus test positive (Investigations) | 0 (0) | 1 (1) | 0 (0)
Thyroxine free decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Transaminases increased (Investigations) | 1 (1) | 2 (2) | 3 (3)
Tri-iodothyronine decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Tri-iodothyronine free decreased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Tri-iodothyronine free increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Troponin I increased (Investigations) | 0 (0) | 1 (1) | 1 (1)
Troponin increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Urine ketone body present (Investigations) | 0 (0) | 1 (1) | 0 (0)
Urine output decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Urine sodium increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Vitamin D decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 39 (42) | 43 (45) | 18 (21)
Weight increased (Investigations) | 4 (4) | 4 (7) | 2 (2)
White blood cell count decreased (Investigations) | 2 (2) | 2 (2) | 19 (33)
White blood cell count increased (Investigations) | 0 (0) | 1 (1) | 2 (3)
Acidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Appetite disorder (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Cachexia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 2 (2)
Decreased appetite (Metabolism and nutrition disorders) | 73 (78) | 89 (101) | 78 (88)
Dehydration (Metabolism and nutrition disorders) | 4 (4) | 10 (11) | 6 (7)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Dyslipidaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0)
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 (0) | 4 (5) | 0 (0)
Failure to thrive (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Fluid imbalance (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Folate deficiency (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Glucose tolerance impaired (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0)
Gout (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hyperalbuminaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hyperamylasaemia (Metabolism and nutrition disorders) | 4 (8) | 0 (0) | 1 (1)
Hypercalcaemia (Metabolism and nutrition disorders) | 6 (7) | 8 (11) | 3 (3)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 3 (3) | 2 (2) | 0 (0)
Hypercreatininaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 11 (13) | 16 (24) | 10 (14)
Hyperkalaemia (Metabolism and nutrition disorders) | 6 (7) | 7 (8) | 7 (8)
Hyperlipasaemia (Metabolism and nutrition disorders) | 1 (4) | 0 (0) | 0 (0)
Hyperlipidaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hypermagnesaemia (Metabolism and nutrition disorders) | 3 (3) | 1 (1) | 0 (0)
Hypernatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1)
Hyperphagia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hyperuricaemia (Metabolism and nutrition disorders) | 6 (8) | 5 (6) | 3 (3)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 9 (10) | 10 (13) | 4 (5)
Hypocalcaemia (Metabolism and nutrition disorders) | 10 (10) | 9 (10) | 7 (9)
Hypochloraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 2 (2) | 4 (4) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 12 (15) | 21 (26) | 16 (17)
Hypomagnesaemia (Metabolism and nutrition disorders) | 3 (4) | 5 (5) | 19 (19)
Hyponatraemia (Metabolism and nutrition disorders) | 9 (10) | 17 (20) | 12 (14)
Hypophagia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 2 (2)
Hypophosphataemia (Metabolism and nutrition disorders) | 5 (5) | 6 (7) | 2 (4)
Hypoproteinaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0)
Hypovolaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Iron deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Malnutrition (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 1 (1)
Metabolic acidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Protein deficiency (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 4 (4) | 5 (5) | 2 (2)
Vitamin D deficiency (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 34 (39) | 24 (27) | 12 (15)
Arthritis (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (3) | 1 (1)
Autoimmune arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Back disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 39 (46) | 38 (45) | 32 (34)
Bone pain (Musculoskeletal and connective tissue disorders) | 5 (5) | 4 (4) | 6 (6)
Bursitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0)
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Clubbing (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Costochondritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Fistula inflammation (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 6 (6) | 8 (10)
Groin pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 3 (3)
Hypertrophic osteoarthropathy (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Joint effusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Joint stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 2 (2)
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 4 (4) | 0 (0)
Limb discomfort (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (2)
Mastication disorder (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Metatarsalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Muscle contracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 5 (6) | 7 (7) | 2 (2)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 6 (6) | 10 (11) | 8 (8)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 16 (16) | 15 (17) | 13 (14)
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 31 (32) | 17 (21) | 7 (7)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 13 (14) | 13 (15) | 16 (30)
Myalgia intercostal (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Myopathy (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Myosclerosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Myositis (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 8 (8) | 11 (12) | 6 (6)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 4 (4) | 1 (1) | 1 (1)
Osteochondrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 19 (21) | 23 (25) | 14 (15)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 1 (1)
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (2)
Periarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Polyarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
SAPHO syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Scleroderma (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Sjogren's syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Soft tissue swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Spinal pain (Musculoskeletal and connective tissue disorders) | 4 (5) | 4 (4) | 0 (0)
Tendon calcification (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Tendon discomfort (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Trismus (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 2 (2) | 2 (2)
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal tract adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Infected neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Oncologic complication (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Pituitary tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Thyroid adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Tumour associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (3) | 2 (3)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 2 (2) | 1 (1)
Tumour thrombosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Ageusia (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Altered state of consciousness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Amnesia (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Aphasia (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Ataxia (Nervous system disorders) | 1 (1) | 2 (2) | 1 (1)
Auditory nerve disorder (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Balance disorder (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Brain oedema (Nervous system disorders) | 1 (1) | 2 (2) | 0 (0)
Carotid artery stenosis (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Carpal tunnel syndrome (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Cerebral infarction (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0)
Cerebral ischaemia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Cognitive disorder (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Disturbance in attention (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Dizziness (Nervous system disorders) | 15 (15) | 25 (35) | 20 (21)
Dizziness postural (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Drooling (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Dysaesthesia (Nervous system disorders) | 1 (1) | 1 (1) | 2 (2)
Dysarthria (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0)
Dysgeusia (Nervous system disorders) | 10 (11) | 8 (8) | 17 (19)
Encephalopathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Facial paralysis (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Head discomfort (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 23 (26) | 25 (36) | 22 (29)
Hemianopia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Horner's syndrome (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0)
Hyperaesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 5 (5) | 8 (11) | 6 (6)
Hypokinesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Intercostal neuralgia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Intracranial aneurysm (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Ischaemic cerebral infarction (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Lethargy (Nervous system disorders) | 3 (3) | 0 (0) | 1 (1)
Loss of consciousness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Memory impairment (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0)
Migraine (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Neuralgia (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0)
Neurological decompensation (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 1 (1) | 5 (5) | 14 (16)
Nystagmus (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 8 (8) | 8 (8) | 14 (15)
Parosmia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Peripheral motor neuropathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1) | 2 (2) | 10 (11)
Peroneal nerve palsy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Polyneuropathy (Nervous system disorders) | 0 (0) | 1 (1) | 12 (12)
Poor quality sleep (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Post herpetic neuralgia (Nervous system disorders) | 0 (0) | 3 (3) | 0 (0)
Radicular syndrome (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Restless legs syndrome (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Sciatica (Nervous system disorders) | 3 (3) | 2 (2) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0)
Seizure like phenomena (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Sensory loss (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Sinus headache (Nervous system disorders) | 0 (0) | 1 (2) | 0 (0)
Somnolence (Nervous system disorders) | 3 (3) | 2 (2) | 0 (0)
Speech disorder (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Spinal cord compression (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Stupor (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 6 (6) | 2 (2) | 2 (2)
Toxic neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Tremor (Nervous system disorders) | 4 (4) | 2 (2) | 3 (3)
Trigeminal neuralgia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Vertebral artery occlusion (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Thrombosis in device (Product Issues) | 1 (1) | 0 (0) | 0 (0)
Adjustment disorder with depressed mood (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Aggression (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Agitation (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 17 (17) | 16 (16) | 9 (9)
Apathy (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0)
Aversion (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Confusional state (Psychiatric disorders) | 5 (5) | 4 (4) | 4 (4)
Delirium (Psychiatric disorders) | 4 (4) | 2 (2) | 1 (1)
Depressed mood (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1)
Depression (Psychiatric disorders) | 3 (3) | 8 (9) | 9 (9)
Disorganised speech (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Disorientation (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Euphoric mood (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Hallucination (Psychiatric disorders) | 0 (0) | 4 (4) | 0 (0)
Hallucination, auditory (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 27 (28) | 37 (42) | 22 (23)
Irritability (Psychiatric disorders) | 1 (1) | 1 (2) | 0 (0)
Libido decreased (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Listless (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Mood altered (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Mood swings (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Nervousness (Psychiatric disorders) | 2 (2) | 0 (0) | 1 (1)
Panic attack (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Panic disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Restlessness (Psychiatric disorders) | 1 (1) | 0 (0) | 2 (2)
Sleep disorder (Psychiatric disorders) | 4 (4) | 2 (2) | 2 (2)
Substance-induced psychotic disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 4 (5) | 5 (5) | 4 (4)
Azotaemia (Renal and urinary disorders) | 1 (1) | 1 (1) | 3 (3)
Bladder dilatation (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Bladder pain (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Chromaturia (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0)
Chronic kidney disease (Renal and urinary disorders) | 0 (0) | 2 (2) | 4 (4)
Dysuria (Renal and urinary disorders) | 2 (2) | 4 (4) | 5 (5)
Glycosuria (Renal and urinary disorders) | 1 (2) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 4 (4) | 5 (7) | 2 (2)
Hydronephrosis (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0)
Leukocyturia (Renal and urinary disorders) | 0 (0) | 2 (2) | 0 (0)
Micturition urgency (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Nephritis (Renal and urinary disorders) | 0 (0) | 2 (2) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Nephropathy toxic (Renal and urinary disorders) | 0 (0) | 0 (0) | 2 (2)
Nocturia (Renal and urinary disorders) | 0 (0) | 6 (6) | 3 (3)
Pollakiuria (Renal and urinary disorders) | 2 (2) | 5 (5) | 3 (3)
Polyuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Prerenal failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Proteinuria (Renal and urinary disorders) | 2 (2) | 7 (7) | 1 (1)
Pyelocaliectasis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 4 (4) | 5 (5)
Renal impairment (Renal and urinary disorders) | 1 (1) | 0 (0) | 2 (3)
Renal pain (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Renal tubular disorder (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Stress urinary incontinence (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Ureteric haemorrhage (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Urethral dilatation (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 2 (2) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 3 (3) | 3 (3) | 2 (2)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 3 (3) | 1 (1) | 1 (1)
Breast enlargement (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Breast pain (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Dyspareunia (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Erectile dysfunction (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 1 (1)
Genital cyst (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Genital rash (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Gynaecomastia (Reproductive system and breast disorders) | 2 (2) | 1 (1) | 0 (0)
Nipple disorder (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Penile haemorrhage (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Penile pain (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Plasma cell balanitis (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Prostatism (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 1 (1)
Scrotal cyst (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Scrotal erythema (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Allergic cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Bronchial secretion retention (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Catarrh (Respiratory, thoracic and mediastinal disorders) | 1 (3) | 0 (0) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 9 (12) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 40 (47) | 38 (41) | 26 (33)
Diaphragmalgia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Dysaesthesia pharynx (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 7 (7) | 4 (4)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 34 (37) | 32 (35) | 31 (35)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 9 (9) | 8 (9) | 5 (5)
Emphysema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 4 (4) | 7 (8)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 8 (8) | 18 (28) | 8 (9)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 1 (1) | 18 (21)
Hyperventilation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2) | 1 (1)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 1 (1)
Laryngeal haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 4 (4) | 3 (3)
Nasal inflammation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Nasal septum deviation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Nasal ulcer (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 7 (8) | 11 (11)
Orthopnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Painful respiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pharyngeal oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 11 (11) | 6 (6) | 5 (5)
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 1 (1)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 1 (1) | 0 (0)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 12 (12) | 2 (2)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 2 (2)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 20 (23) | 23 (26) | 18 (18)
Pulmonary artery thrombosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 5 (5) | 2 (2)
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2) | 0 (0)
Pulmonary pain (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 1 (1)
Respiratory acidosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Restrictive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 2 (2)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 8 (9) | 8 (10) | 11 (11)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Sputum increased (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Sputum retention (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 1 (1)
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Throat tightness (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 0 (0)
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2) | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2)
Actinic keratosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 3 (4) | 8 (9) | 42 (42)
Angioedema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Blister (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 1 (1)
Butterfly rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Chloasma (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Cold sweat (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (2)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 4 (4) | 3 (3) | 5 (5)
Dermal cyst (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 3 (3) | 1 (1) | 0 (0)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 3 (4) | 4 (5) | 0 (0)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Drug eruption (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (3) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 16 (17) | 21 (22) | 7 (7)
Ecchymosis (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 4 (4) | 4 (4) | 1 (1)
Eczema asteatotic (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 6 (6) | 4 (6) | 3 (3)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2) | 0 (0)
Exfoliative rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Haemorrhage subcutaneous (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Hair growth abnormal (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 4 (4) | 6 (6) | 3 (3)
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2) | 0 (0)
Intertrigo (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Koilonychia (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Lichenoid keratosis (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Macule (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) | 0 (0)
Milia (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Miliaria (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Nail dystrophy (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 4 (4) | 5 (5) | 2 (2)
Nodular vasculitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Onycholysis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Onychomadesis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Pain of skin (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Papule (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0)
Penile ulceration (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Petechiae (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3) | 0 (0)
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Pigmentation disorder (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Post inflammatory pigmentation change (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 42 (53) | 67 (81) | 17 (21)
Pruritus generalised (Skin and subcutaneous tissue disorders) | 2 (2) | 3 (3) | 1 (1)
Psoriasis (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 39 (49) | 57 (66) | 40 (44)
Rash erythematous (Skin and subcutaneous tissue disorders) | 3 (3) | 1 (1) | 0 (0)
Rash generalised (Skin and subcutaneous tissue disorders) | 4 (4) | 2 (2) | 1 (1)
Rash macular (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 10 (10) | 20 (22) | 2 (2)
Rash papular (Skin and subcutaneous tissue disorders) | 1 (2) | 2 (2) | 0 (0)
Rash pruritic (Skin and subcutaneous tissue disorders) | 2 (2) | 3 (3) | 0 (0)
Rash vesicular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Scab (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Skin discolouration (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Skin exfoliation (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0) | 2 (6)
Skin fissures (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Skin induration (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Skin irritation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Skin lesion (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2) | 0 (0)
Skin mass (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3) | 0 (0)
Skin necrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Skin swelling (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 1 (1)
Swelling face (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 2 (2)
Toxic skin eruption (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 6 (6) | 3 (5) | 5 (5)
Vitiligo (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 1 (1)
Angiopathy (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Arterial thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Brachiocephalic vein occlusion (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Capillary leak syndrome (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Circulatory collapse (Vascular disorders) | 1 (1) | 1 (3) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 4 (4) | 6 (6)
Embolism (Vascular disorders) | 0 (0) | 3 (3) | 4 (5)
Flushing (Vascular disorders) | 0 (0) | 2 (2) | 2 (2)
Haematoma (Vascular disorders) | 1 (1) | 2 (2) | 1 (1)
Hot flush (Vascular disorders) | 0 (0) | 0 (0) | 4 (4)
Hyperaemia (Vascular disorders) | 1 (1) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 17 (18) | 16 (19) | 5 (5)
Hypertensive crisis (Vascular disorders) | 0 (0) | 1 (2) | 0 (0)
Hypotension (Vascular disorders) | 7 (7) | 6 (6) | 8 (10)
Ischaemic limb pain (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Jugular vein distension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Microangiopathy (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 1 (1) | 2 (2)
Pallor (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Peripheral arterial occlusive disease (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Peripheral ischaemia (Vascular disorders) | 0 (0) | 1 (1) | 1 (1)
Phlebitis (Vascular disorders) | 0 (0) | 1 (1) | 6 (7)
Superior vena cava occlusion (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Superior vena cava syndrome (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Thrombophlebitis (Vascular disorders) | 2 (2) | 0 (0) | 2 (2)
Thrombophlebitis superficial (Vascular disorders) | 0 (0) | 2 (2) | 1 (1)
Thrombosis (Vascular disorders) | 0 (0) | 2 (2) | 1 (1)
Varicose vein (Vascular disorders) | 0 (0) | 0 (0) | 3 (3)
Vasculitis (Vascular disorders) | 1 (1) | 0 (0) | 1 (1)
Vasoconstriction (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Vasodilatation (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Vein disorder (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Venous thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2018-01-09): https://cdn.clinicaltrials.gov/large-docs/82/NCT02453282/Prot_015.pdf
  • Statistical Analysis Plan (2017-06-20): https://cdn.clinicaltrials.gov/large-docs/82/NCT02453282/SAP_000.pdf